# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for DMID Protocol: 19-0015

**Study Title:** 

Mucosal immune responses against *Neisseria gonorrhoeae* following meningococcal immunization in healthy young adults

NCT04722003

Version 1.0

**DATE: 22NOV2023** 

RESTRICTED

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 19-0015 |
|---|---|
| Protocol Version: | 7.0 |
| <b>Development Phase:</b> | Phase II |
| Products: | Bexsero® (4CMenB), FDA-approved multi-component meningococcal serogroup B vaccine |
| Form/Route: | Intramuscular injection |
| <b>Indication Studied:</b> | Neisseria gonorrhoeae |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | July 19, 2021 |
| <b>Clinical Trial Completion Date:</b> | October 2, 2023 |
| Date of the Analysis Plan: | November 22, 2023 |
| Version Number: | V1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | 2 |
|---|---|---|
| TABLE | OF CONTENTS | 3 |
| LIST O | F ABBREVIATIONS | 6 |
| 1. | PREFACE | 9 |
| 2. | INTRODUCTION | 10 |
| 2.1. | Purpose of the Analyses | 11 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 12 |
| 3.1. | Study Objectives | 12 |
| 3.1.1. | Primary Objective | 12 |
| 3.1.2. | Secondary Objective | 12 |
| 3.1.3. | Exploratory Objectives | 12 |
| 3.2. | Endpoints | 12 |
| 3.2.1. | Primary Outcome | 12 |
| 3.2.2. | Secondary Outcomes | 13 |
| 3.2.3. | Exploratory Outcomes | 13 |
| 3.3. | Study Definitions and Derived Variables | 14 |
| 3.3.1. | Baseline Values | 14 |
| 3.3.2. | Immunogenicity Outcomes | 14 |
| 4. | INVESTIGATIONAL PLAN | 16 |
| 4.1. | Overall Study Design and Plan | 16 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 16 |
| 4.3. | Selection of Study Population | 16 |
| 4.4. | Treatments | 16 |
| 4.4.1. | Treatments Administered. | 16 |
| 4.4.2. | Identity of Investigational Product(s) | 17 |
| 4.4.3. | Method of Assigning Participants to Treatment Groups (Randomization) | 17 |
| 4.4.4. | Selection and Timing of Dose for Each Participant | 17 |
| 4.4.5. | Blinding | 17 |
| 4.4.6. | Prior and Concomitant Therapy | 18 |
| 4.4.7. | Treatment Compliance | 18 |
| 4.5. | Immunogenicity and Safety Variables | 18 |

# Table of Contents (continued)

| 4.5.1. | Immunogenicity Variables | 18 |
|--------|--------------------------------------------------|----|
| 4.5.2. | Safety Variables | 19 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 20 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 21 |
| 6.1. | General Principles | 21 |
| 6.2. | Timing of Analyses | 21 |
| 6.3. | Analysis Populations | 21 |
| 6.3.1. | Immunogenicity Populations | 21 |
| 6.3.2. | Per Protocol (PP) Populations for Immunogenicity | 22 |
| 6.3.3. | Safety Population | 22 |
| 6.4. | Covariates and Subgroups | 22 |
| 6.5. | Missing Data | 22 |
| 6.6. | Interim Analyses and Data Monitoring | 22 |
| 6.7. | Multiple Comparisons/Multiplicity | 23 |
| 7. | STUDY PARTICIPANTS | 24 |
| 7.1. | Disposition of Participants | 24 |
| 7.2. | Protocol Deviations | 24 |
| 8. | IMMUNOGENICITY EVALUATION | 25 |
| 8.1. | Primary Outcome Analysis | 25 |
| 8.2. | Secondary Outcome Analyses | 25 |
| 8.3. | Exploratory Outcome Analyses | 25 |
| 9. | SAFETY EVALUATION | 27 |
| 9.1. | Demographic and Other Baseline Characteristics | 27 |
| 9.1.1. | Pre-Existing Medical Conditions | 27 |
| 9.1.2. | Prior and Concomitant Medications | 27 |
| 9.2. | Measurements of Treatment Compliance | 27 |
| 9.3. | Adverse Events | 27 |
| 9.3.1. | Solicited Events and Symptoms | 28 |
| 9.3.2. | Unsolicited Adverse Events. | 28 |
| 9.4. | Pregnancies | 29 |
| 9.5. | Clinical Laboratory Evaluations | 29 |
| 9.6. | Vital Signs | 29 |

# Table of Contents (continued)

| 9.7. | Physical Examinations | 29 |
|-------|----------------------------------------------------------|-----|
| 9.8. | Concomitant Medications | 30 |
| 9.9. | Other Safety Measures | 30 |
| 10. | OTHER ANALYSES | 31 |
| 11. | REPORTING CONVENTIONS | 32 |
| 12. | TECHNICAL DETAILS | 33 |
| 13. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STU<br>ANALYSES | |
| 14. | REFERENCES | 35 |
| 15. | LISTING OF TABLES, FIGURES, AND LISTINGS | 37 |
| APPEN | DICES | 38 |
| APPEN | DIX 1. TABLE MOCK-UPS | 39 |
| APPEN | DIX 2. FIGURE MOCK-UPS | 107 |
| APPEN | DIX 3. LISTINGS MOCK-UPS | 129 |

# LIST OF ABBREVIATIONS

| 4CMenB | Bexsero® or multi-component meningococcal serogroup B vaccine |
|---|---|
| ACIP | Advisory Committee on Immunization Practices |
| AE | Adverse Event/Adverse Experience |
| aPTT | Activated Partial Thromboplastin Time |
| BLA | Biologics License Applications |
| BMI | Body Mass Index |
| CI | Confidence Interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| COVID-19 | Coronavirus disease 2019 |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| СТ | Chlamydia trachomatis |
| DCC | Data Coordinating Center |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-Linked Immunosorbent Assay |
| FDA | Food and Drug Administration |
| FHbp | factor H binding protein |
| GC | Neisseria gonorrhoeae |
| GC | Good Clinical Practice |
| GMFR | Geometric Mean Fold Rise |
| GMT | Geometric Mean Titer |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | Human Immunodeficiency Virus |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| ICS | Intracellular Cytokine Staining |
| IDCRC | Infectious Diseases Clinical Research Consortium |
| IDES | Internet Data Entry System |
| IgA | Immunoglobin A |
| IgG | Immunoglobin G |
| IM | Intramuscular |
| IND | Investigational New Drug Application |

# List of Abbreviations (continued)

| IRB | Institutional Review Board |
|--------|------------------------------------------------------------------|
| ISM | Independent Safety Monitor |
| IUD | Intrauterine Device |
| JAMA | Journal of the American Medical Association |
| LLC | Limited Liability Corporation |
| MAAEs | Medically-Attended Adverse Events |
| MBC | Memory B Cell |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MeNZB | New Zealand Meningococcal Group B Vaccine |
| mL | Milliliter |
| mm | Millimeter |
| N | Number (typically refers to participants) |
| NAAT | Nucleic Acid Amplification Test |
| NadA | Neisserial Adhesion A |
| NHBA | Neisserial Heparin Binding Antigen |
| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
| NIH | National Institutes of Health |
| NSAID | Non-Steroidal Anti-Inflammatory Drug |
| OMV | Outer Membrane Vesicle |
| PBMC | Peripheral Blood Mononuclear Cell |
| PI | Principal Investigator |
| PID | Pelvic Inflammatory Disease |
| PL | Platelet Count |
| PorA | Porin protein |
| PP | Per Protocol |
| PT | Prothrombin Time |
| RPR | Rapid Plasma Regain |
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SAP | Statistical Analysis Plan |
| SBA | Serum Bactericidal Antibody |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| STI | Sexually Transmitted Infection |
| USP | United States Pharmacopeial Convention |
| VTEU | Vaccine and Treatment Evaluation Unit |

# List of Abbreviations (continued)

| WBC | White Blood Count |
|-----|---------------------------|
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "Mucosal immune responses against Neisseria gonorrhoeae following meningococcal immunization in healthy young adults" (DMID Protocol 19-0015) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. A separate report shell will be created for the interim immunogenicity analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice. This SAP also follows the FDA guidance regarding the COVID-19 public health emergency. 1. Contingency measures implemented to manage study conduct during disruption of the study as a result of COVID-19 control measures. 2. All participants affected by the COVID-19 will be highlighted. 3. Analyses and corresponding discussions that address the impact of implemented contingency measures. 4. Any protocol deviation due to COVID-19 will be documented.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3). Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Gonorrhea is a sexually transmitted infection (STI) caused by the gram-negative diplococcus *Neisseria* gonorrhoeae (GC). In 2012 the World Health Organization (WHO) estimated approximately 78 million new cases of gonorrhea globally[1]. In the United States, gonorrhea is the second most reported notifiable disease, with more than 550,000 cases reported in 2017. Rates of gonococcal disease have been steadily increasing since 2009 irrespective of age, sex, ethnic group, or geographic region.

Though gonococcal infections are curable with antibiotic therapy, antimicrobial resistance has become a global public health problem. The prevalence of resistance to multiple antibiotic classes has increased gradually since the 1940s,[1] and GC isolates with reduced susceptibility to current first-line therapy – ceftriaxone and azithromycin – have emerged.[2] Given the large and growing burden of disease, and the threat of untreatable gonococcal infections due to antimicrobial resistance, a safe and effective vaccine is urgently needed. Unfortunately, previous efforts to develop a gonorrhea vaccine have been largely unsuccessful.

Recently, a retrospective case-control study in New Zealand demonstrated 31% (95% confidence interval (CI), 21-39) effectiveness of an outer membrane vesicle (OMV) meningococcal group B vaccine (MeNZB) against incident gonorrhea.[3] The same group of investigators also reported 24% (95% CI, 1-42) vaccine effectiveness against hospitalization caused by gonorrhea.[3] Previous ecological studies had suggested a possible protective effect of OMV vaccines against gonorrhea in Norway[4] and Cuba.[5] Meningococcal OMV vaccines have been used successfully to control epidemic strains of *N. meningitidis* serogroup B.[6] These vaccines elicit serum bactericidal antibody (SBA) responses directed primarily against meningococcal strain-specific porin protein, PorA.[7] The precise mechanism of cross-protection conferred by meningococcal OMV vaccines against GC remains unknown.

A four component meningococcal serogroup B vaccine (Bexsero® or 4CMenB) was recently licensed for use in the United States and was given a category B recommendation by the Advisory Committee on Immunization Practices (ACIP) for use in adolescents and young adults aged 10- 25 years,[8] which is administered intramuscularly as a two dose-series, with the second dose given at least one month after the first dose.

4CMenB includes OMVs containing PorA serosubtype P1.4, as well as three recombinant protein antigens (neisserial adhesion A [NadA], factor H binding protein [FHbp] fusion protein, and neisserial heparin binding antigen [NHBA] fusion protein).[9] An analysis of gonococcal incidence following a 4CMenB vaccination campaign in one region of Quebec, Canada found a non-significant reduction in gonorrhea cases in the post-vaccination period,[10] supporting the findings from New Zealand, and suggesting that 4CMenB vaccine could protect against gonorrhea.

A recent study found a high level of amino acid sequence identity between the 4CMenB OMV antigens and those in the MeNZB OMV in the vaccine studied in New Zealand, and with OMV homologues in a laboratory strain of GC. The same study found that rabbits vaccinated either with MeNZB or the OMV component of 4CMenB raised antibodies against GC, and that 4CMenB vaccination in humans elicited serum antibodies against GC.[11] In contrast, another study found vaccination with a native OMV vaccine raised SBA responses against GC in mice, but 4CMenB vaccination did not elicit similar SBA responses in humans.[12]

Given the potential public health impact of an effective vaccine against gonorrhea, a better understanding of the immunologic responses to GC following 4CMenB vaccination is needed. Specifically, although two studies have characterized antibody responses against GC following 4CMenB in serum, gonorrhea is a mucosal disease. While there are studies looking at the ability of meningococcal serogroup B vaccines to

modulate human nasopharyngeal mucosal immunity to *N. meningitidis*, there are no data on the impact of 4CMenB on immunologic responses at the human mucosal surfaces where GC is typically encountered (urethra, rectum, cervix, and pharynx).

This is a mechanistic clinical trial to assess the systemic and mucosal immunogenicity of the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against GC, using a placebo vaccine (normal saline) as a comparator, in healthy young adults.

# 2.1. Purpose of the Analyses

These analyses will assess the immunogenicity and safety of the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against GC in comparison with a placebo vaccine (normal saline) and will be included in the clinical study report.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

# 3.1.1. Primary Objective

• To characterize the rectal mucosal IgG antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine (normal saline) in healthy adult participants.

#### 3.1.2. Secondary Objective

- To characterize the serum IgG antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To assess the safety and reactogenicity of 4CMenB in healthy adult participants.

# 3.1.3. Exploratory Objectives

- To characterize the vaginal mucosal IgG antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To characterize the oropharyngeal mucosal IgG antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants
- To characterize the serum IgA antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To characterize the mucosal IgA antibody response to GC elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants
- To characterize the systemic B cell responses to GC antigens elicited by 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To characterize the systemic T cell responses to GC antigens elicited by 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To characterize the mucosal T cell responses to GC antigens elicited by 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To characterize the serum bactericidal antibody responses to GC elicited by 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants.
- To evaluate the impact of 4CMenB vaccine-induced antibodies on gonococcal adhesion to human cervical cells.
- To characterize immune responses to *N. meningitidis* elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult participants for use as controls.

# 3.2. Endpoints

#### 3.2.1. Primary Outcome

• Rectal mucosal IgG concentrations (geometric mean titers, GMT) against GC OMV antigens at Day 1, 29, 43, 57, and 181 in each treatment group.

#### 3.2.2. Secondary Outcomes

- Serum IgG concentrations (GMT) against GC OMV antigens at Day 1, 29, 43, 57, and 181 in each treatment group
- Frequency and severity of any AE related to 4CMenB immunization through the end of the study.
- Frequency of SAEs through the end of the study.

#### 3.2.3. Exploratory Outcomes

- Rectal mucosal IgG concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Serum IgG concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Vaginal mucosal IgG concentrations geometric mean titer (GMT) against GC antigens before and after vaccination in female participants in each treatment group
- Oropharyngeal mucosal IgG concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Serum IgA concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Rectal mucosal IgA concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Vaginal mucosal IgA concentrations (GMT) against GC antigens before and after vaccination in female participants in each treatment group
- Oropharyngeal mucosal IgA concentrations (GMT) against GC antigens before and after vaccination in each treatment group
- Frequencies and function of memory B cells specific for antigens from GC before and after vaccination by ELISpot in each treatment group.
- Frequencies and function of peripheral blood T cells specific for antigens from GC before and after vaccination by ELISpot in each treatment group.
- Frequencies, phenotype, and function of peripheral blood CD4+ T cells specific for antigens from GC based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.
- Frequencies, phenotype, and function of peripheral blood CD8+ T cells specific for antigens from GC based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.
- Frequencies, phenotype, and function of rectal mucosal CD4+ T cells specific for antigens from GC based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.
- Frequencies, phenotype, and function of rectal mucosal CD8+ T cells specific for antigens from GC based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.

- Serum bactericidal antibody titers against GC before and after vaccination in each treatment group.
- Percent inhibition of gonococcal adhesion to human cervical cell line (ME180) by mucosal antibodies at Day 43 in each treatment group.
- Serum IgG concentrations (GMT) against *N. meningitidis* antigens before and after vaccination in each treatment group.
- Frequencies and function of memory B cells specific for antigens from *N. meningitidis* before and after vaccination by ELISpot in each treatment group.
- Frequencies and function of peripheral blood T cells specific for antigens from *N. meningitidis* before and after vaccination by ELISpot in each treatment group.
- Frequencies, phenotype, and function of peripheral blood CD4+ T cells specific for antigens from *N. meningitidis* based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.
- Frequencies, phenotype, and function of peripheral blood CD8+ T cells specific for antigens from *N. meningitidis* based on cytokine profile before and after vaccination by intracellular cytokine staining in each treatment group.

# 3.3. Study Definitions and Derived Variables

#### 3.3.1. Baseline Values

The baseline value will be defined as the last value obtained prior to the first vaccination/dose of study product. The Immunogenicity baseline for serum, mucosal secretion (vaginal, rectal and oropharyngeal) sample will be taken at enrollment day (Visit 01) and rectal mucosal biopsy baseline will be taken at visit 00C, which is 14 - 28 days before enrollment.

#### 3.3.2. Immunogenicity Outcomes

In the primary, secondary, and exploratory outcomes, the GMT for Enzyme-Linked Immunosorbent Assay (ELISA) will be calculated for Days 1, 29, 43, 57 and 181 for each treatment arm. The GMT is defined as:

$$GMT = \sqrt[n]{X1 * X2 * X3 * ... ... * Xn}$$

In practice, it is the equivalent of:  $GMT = Exp\{[log(X1) + log(X2) + ... + log(Xn)] / n\}$ 

Where the X1, X2, ...Xn are the titers for each participant at a certain timepoint. A sample SAS code for calculating the geometric mean and the 95% confidence interval is shown below.

proc surveymeans data=data geomean; var variable; run;

The geometric mean fold rise (GMFR) for ELISA titers will be calculated for Days 29, 43, 57, and 181 compared to baseline titer in each study arm. The fold change for each participant at each timepoint is calculated first by dividing the follow-up titer by the baseline titer, then the geometric mean and 95% confidence interval will be calculated for each treatment arm at each timepoint.

Similarly, the ratio of serum to mucosal (rectal, vaginal, and oropharyngeal) IgG will be calculated at each time point. The geometric mean and confidence interval will be calculated as above.

Percent inhibition of gonococcal adhesion to human cervical cell line by mucosal antibody is defined as:

100% \* [(Titer without mucosal antibody – Titer with mucosal antibody) / Titer without mucosal antibody]

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a single site, phase 2, double blinded, mechanistic clinical trial to assess the systemic and mucosal immunogenicity of the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against *N. gonorrhoeae* (GC), using a placebo vaccine (normal saline) as a comparator. Approximately 50 participants (maximum of 60 participants) who meet all eligibility criteria will be randomized 4:1 to one of two treatment groups. Group 1 (approximately N=40) will receive two doses of 4CMenB on Day 1 and Day 29. Group 2 (approximately N=10) will receive two placebo injections on Day 1 and Day 29. Both treatment groups include a rectal mucosal biopsy cohort and a no rectal biopsy cohort, and the participants in each cohort will be stratified by sex. The goal will be to ensure adequate representation of participants by sex in both groups (see **Table 1**).

Potential participants will be screened for eligibility during the screening visit(s). Informed consent will be obtained. All participants undergo a brief medical history and sexual history, a concomitant medication review, a directed physical examination, STI screening, etc. See the protocol for detailed eligibility criteria.

The screening/enrollment period will be approximately 6 months and participants will be followed through 6 months after their first vaccination. The duration of each participant's participation is approximately 8 months, from recruitment through the last study visit.

This clinical study will utilize a Safety Monitoring committee (SMC), which is an independent group of experts that advises the DMID. The primary responsibility of the SMC is to monitor participant safety.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

This study follows a double-blind, randomized, placebo concurrent control design. Participants receive either the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against GC or saline placebo as their first study vaccination. After approximately 1 month, all participants will receive the second dose of study vaccine (or placebo). To date, there are no vaccines that are licensed in preventing gonorrhea, thus a placebo will be used as the comparator, which allows us to determine if the observed effects are due to the study product or other reason.

# **4.3.** Selection of Study Population

The study population will include approximately 50 males and non-pregnant females, 18 to 49 years of age, inclusive, who are in good health and meet all eligibility criteria. Participants will be recruited from the community at large and enrolled at 1 VTEU site (Hope Clinic, Emory VTEU). This age range was selected to represent the population with the highest incidence of gonorrhea therefore children are excluded from this study. There are no plans currently to include children in future studies of mucosal immune responses to GC after meningococcal immunization.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

The multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against GC or saline placebo as study vaccination at day 1 and 29.

# 4.4.2. Identity of Investigational Product(s)

Bexsero or 4CMenB: Active Product. Each 0.5-mL dose of Bexsero (4CMenB) is formulated to contain 50 micrograms each of recombinant proteins NadA, NHBA, and fHbp, 25 micrograms of OMV, 1.5 mg aluminum hydroxide (0.519 mg of Al3+), 3.125 mg sodium chloride, 0.776 mg histidine, and 10 mg sucrose at pH 6.4 – 6.7. The NadA component is a fragment of the full-length protein derived from *N. meningitidis* strain 2996 (peptide 8 variant 2/3). The NHBA component is a recombinant fusion protein comprised of NHBA (peptide 2) and accessory protein 953 derived from *N. meningitidis* strains NZ98/254 and 2996, respectively. The fHbp component is a recombinant fusion protein comprised of fHbp (variant 1.1) and the accessory protein 936 derived from *N. meningitidis* strains MC58 and 2996, respectively. These 3 recombinant proteins are individually produced in *Escherichia coli* and purified through a series of column chromatography steps. The OMV antigenic component is produced by fermentation of *N. meningitidis* strain NZ98/254 (expressing outer membrane protein PorA serosubtype P1.4), followed by inactivation of the bacteria by deoxycholate, which also mediates vesicle formation. The antigens are adsorbed onto aluminum hydroxide. Each dose contains less than 0.01 micrograms kanamycin (by calculation).

Placebo: The placebo is 0.9% Sodium Chloride, USP injection.

#### 4.4.3. Method of Assigning Participants to Treatment Groups (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system, maintained by the Statistical and Data Coordinating Center (SDCC).

This study will enroll both male and non-pregnant female participants. The goal will be to ensure approximately adequate representation of participants by sex in both Treatment groups (**Table 1**). To facilitate this, randomization will be stratified by sex. Within each biopsy cohort (Rectal Mucosal Biopsy Cohort and No Rectal Mucosal Biopsy Cohort), participants will be randomized 4:1 to 4CMenB or placebo. Approximately twenty (20) participants, 10 males and 10 females, will be enrolled into the Rectal Mucosal Biopsy Cohort and approximately 30 participants, 15 males and 15 females, will be enrolled into the No Rectal Mucosal Biopsy Cohort.

The list of randomized treatment assignments will be included in the enrollment module of Emmes' Internet Data Entry System (IDES). Advantage eClinical® will assign each enrolled participant to a treatment arm after demographic and eligibility data have been entered into the system. A designated individual at the site will be provided with a coded list for emergency unblinding purposes, which will be kept in a secure place.

Participant Inclusion and Exclusion Criteria (Section 5.1 of the protocol) must be confirmed by a study clinician licensed to make medical diagnoses and listed on the Form FDA 1572 as the site principal investigator (PI) or sub-investigator. No exemptions are granted on Participant Inclusion/Exclusion Criteria in DMID sponsored studies. Questions about eligibility will be directed toward the DMID Medical Officer.

#### 4.4.4. Selection and Timing of Dose for Each Participant

Bexsero (4CMenB) or placebo will be administered as a 2-dose series (0.5-mL each) in participants randomized to each treatment arm. Both treatment arms will be enrolled and receive the first dose at day 1 (Visit 01) and will receive second dose at day 29 (Visit 04).

#### 4.4.5. Blinding

This is a double-blinded clinical trial. Participants, site investigators, and study personnel who perform study assessments following study product administration, data entry personnel at the sites, and laboratory personnel performing study assays will be blinded to treatment assignment. Syringes will be labeled with an

overlay/blinding tape containing the participant ID, and the treatment number from the treatment key, and expiration time for the syringe, and provided to the unblinded vaccine administrator. The unblinded vaccine administrator will be credentialed to administer vaccines but will not be involved in study-related assessments, participant contact, or data collection following vaccination.

The SMC may receive data in aggregate and presented by study arm. The SMC may be unblinded to individual study treatment assignments, as needed, to adequately assess safety issues. The SMC will review grouped and unblinded data in the closed session only.

# 4.4.6. Prior and Concomitant Therapy

Concomitant medications will include all current medications and non-study vaccinations taken within 30 days before signing the ICF through approximately 28 days after the last study vaccination, and for new-onset chronic medical conditions through the final study visit for each participant. Participants who do not receive all vaccinations will have concomitant medications collected through approximately 28 days after the last vaccination, or early termination, whichever occurs first. Prescription and over-the-counter drugs will be included as well as herbals, vitamins, and supplements. See Section 7.1.2 of the study protocol for more detail.

# 4.4.7. Treatment Compliance

All participants are to receive two doses of either the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero) against GC or saline placebo as their study vaccination at day 1 and 29. Treatment compliance with study product will be defined as the participant receiving all assigned doses within the assigned visit windows. A participant is not in compliance with the protocol treatment if they miss at least one dose or receive at least one dose out of the visit window. When this happens, it will be recorded as a protocol deviation, and the participant will be excluded from the per-protocol population (Section 6.3.2).

# 4.5. Immunogenicity and Safety Variables

#### 4.5.1. Immunogenicity Variables

See **Table 2** for the schedule of study procedures.

Immunogenicity testing will include antibody assays, cell-mediated immunity assays, and bacterial adhesion assays. Antibody assays will be performed to measure the IgG and IgA concentrations against GC antigens at mucosal sites (rectum, vagina, oropharynx) and in serum, serum IgG concentrations against N. meningitidis antigens by enzyme-linked immunosorbent assay (ELISA), and serum bactericidal antibody titers determined by assessing GC survival in the presence of a fixed concentration of human complement source and serially diluted sera in which complement has been heat inactivated. Cell-mediated immunity assays will be performed to measure frequencies and function of memory B cells (MBC) and peripheral blood T cells specific for GC and N. meningitidis antigens by ELISpot. Cell-mediated immunity assays will be performed to measure frequencies, phenotype and function of peripheral blood CD4+ and CD8+ T cells and rectal mucosal CD4+ and CD8+ T cells specific for GC antigens by intracellular cytokine staining (ICS). Similar assays will also be performed with peripheral blood CD4+ and CD8+ T cells specific for N. meningitidis antigens. A bacterial adhesion assay will be performed to measure the percent inhibition by mucosal antibodies of gonococcal adhesion to a ME180 human cervical cell line at Day 43 in each treatment group. Serum for systemic immunity assays will be collected at days 1 (pre-vaccination), 8, 15, 29, 36, 43, 57 and 181. Serum and mucosal (rectum, vagina, oropharynx) samples for antibody assays will be collected at days 1 (pre-vaccination), 29, 43, 57 and 181.

The immunogenicity variables are:Concentration of mucosal antibodies (IgG or IgA) against GC antigens at mucosal sites (rectum, vagina oropharynx) and serum antibodies (IgG or IgA) against GC antigens. These will be measured by ELISA from specimens collected at each visit (days 1, 29, 43, 57 and 181), and results will be reported as geometric mean titer and 95% confidence interval for each time point for the two treatment arms.

- Frequencies and function of memory B cells and T cells from peripheral blood for GC and *N. meningitidis* antigens will be measured at each visit with ELISpot. The frequencies (cell count) will be reported. Frequencies and function of CD4+ and CD8+ T cells specific for GC and *N. meningitidis* antigens from peripheral blood, and GC antigens from rectal mucosae. These will be measured at each visit with ICS. Cell frequencies will be reported.
- Serum bactericidal antibody against GC and *N. meningitidis* will be measured and reported as geometric mean titer and 95% confidence interval for each time point for the two treatment arms.
- Inhibition of bacterial adhesion to a human cervical cell line (ME180) by mucosal antibodies will be measured by bacterial adhesion assay, and geometric mean titer and 95% confidence interval at each time point for two treatment arms will be reported.
- Other exploratory Immunogenicity outcomes measured by ELISA, ELISpot, and bacterial adhesion assays will be reported similarly.

#### 4.5.2. Safety Variables

Safety will be assessed throughout the study.

Reactogenicity will be measured by pre-vaccination reactogenicity assessment, evaluation of the vaccination site and AE/SAEs from the clinic and self-reported reactogenicity information in an electronic memory aid with a paper back up.

Safety will be assessed by the frequency and severity of any AE related to 4CMenB immunization through the end of the study, and any SAEs through the end of the study.

#### 5. SAMPLE SIZE CONSIDERATIONS

A total of approximately 50 participants (maximal 60) will be enrolled and randomized to one of two study arms, 40 participants will be randomized to the 4CMenB arm and 10 participants to the placebo arm. The 4:1 allocation ratio was not selected based on any formal statistical criteria but instead was selected to maximize the number of participants administered 4CMenB, and thus maximize the amount of immunogenicity data collected on participants administered 4CMenB. Of the 50 participants, 20 participants will be enrolled into the Rectal Mucosal Biopsy Cohort. As with the overall sample size, this number was not selected based on any statistical criteria but was selected weighing the feasibility of enrolling participants who would consent to the biopsy procedure against ensuring ample data was collected via rectal mucosal biopsy as there are no data on the impact of 4CMenB on immunologic responses at the human mucosal surfaces where GC is typically encountered.

This study is not designed to formally test any hypotheses associated with the safety or immunogenicity data.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

Unless otherwise specified, continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, minimum and maximum. For some immunogenicity outcomes, the titers /frequencies will be summarized by geometric mean titer (GMT) /geometric mean titer frequencies and confidence interval (CI), fold change (rise or decline) from baseline will be calculated for the follow up immunogenicity outcomes. When calculating geometric mean, only non-zero values will be included. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. Exact confidence intervals for binomial proportions will be computed for safety variables. In general, all data will be listed, sorted by Treatment group, and participant, and when appropriate by visit number within participant. All summary tables will be structured with a column for each Treatment in the order presented and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

# **6.2.** Timing of Analyses

There will be an interim immunogenicity analysis, which may be used to optimize and prioritize research laboratory assays for exploratory outcomes. The interim immunogenicity analysis will include all available antibody data for the first 20 participants who complete Visit 6, which includes data addressing the primary and secondary objectives, as well as several exploratory objectives.

The final analysis will be performed when all enrolled participants have completed the day 181 visit, the clinical database has been cleaned, monitored, and locked, and data is available for all secondary immunogenicity measures. Exploratory immunogenicity assays will be determined and performed pending the results of the interim immunogenicity analysis. The results for primary and secondary endpoints, including safety data, will be reported in the primary Clinical Study Report (CSR). A CSR addendum will be prepared to report the results for exploratory endpoints and any additional results.

# 6.3. Analysis Populations

Demographic and baseline characteristics will be presented for all enrolled participants. All safety summaries will be presented for the safety population. Immunogenicity measures will be presented for the Immunogenicity and per protocol (PP) populations. A tabular listing of all participants, visits, and observations excluded from analyses will be provided in the CSR.

# **6.3.1.** Immunogenicity Populations

For the primary outcome analysis, the immunogenicity population at a specified follow-up visit will include all eligible participants who have received all doses of study product prior to that visit and have immunogenicity data available for that visit. For this study the Immunogenicity population includes all participants who received at least one dose of study vaccine and contributed at least one sample for immunogenicity testing for which valid results were reported. To account for participants having data available only for a subset of assays, assay-specific populations will be defined. For example, the assays for vaginal mucosal specimens will only include female participants in the immunogenicity population, and rectal mucosal biopsy assays will only include biopsy cohort participants in the immunogenicity population. The population is defined for the participant at baseline, such that even when there is a missing value at a certain follow up visit, the participant will be included in the immunogenicity population.

For analyses using the Immunogenicity population, participants will be classified according to the study product received.

#### 6.3.2. Per Protocol (PP) Populations for Immunogenicity

Per-protocol populations will be defined that further restrict the immunogenicity analysis populations to exclude participants with major protocol deviations or events that may impact study product effectiveness or the ascertainment or interpretation of assay results. The per protocol (PP) population includes all participants in the Immunogenicity subset with the following exclusions: 1) Data from all available visits for participants found to be ineligible at baseline or during follow-up. 2) Data from all visits subsequent to major protocol deviations, such as: a) at least one dose of study vaccination not received; b) at least one dose of study vaccination received at > 4 days out of window.

#### 6.3.3. Safety Population

The safety analysis population includes all participants who received at least one dose of study treatment. For analyses using the safety population, participants will be grouped by study treatment received.

# 6.4. Covariates and Subgroups

Randomization was stratified by sex; however, the protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

# 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If such data points are identified as scientifically valid outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

If a participant missed visits, discontinued vaccinations or early terminated due to Covid-19, the participant will be recorded and highlighted in the report.

# 6.6. Interim Analyses and Data Monitoring

There will be an interim immunogenicity analysis, which may be used to optimize and prioritize research laboratory assays for exploratory outcomes. Results of the interim analyses will not be used to make any decisions concerning the conduct of this trial.

The interim immunogenicity analysis will include all available antibody data for the first 20 participants who complete Visit 6, which includes data addressing the primary and secondary objectives, as well as several exploratory objectives. The interim report will be prepared by the unblinded statistician at the SDCC after all relevant immunogenicity data through Visit 6 are received. Results will be shared only with relevant study personnel (i.e. PI, laboratory investigator(s), and DMID) and only in aggregate by treatment arm. Study personnel will remain blinded to individual participant treatment assignments.

The interim immunogenicity analyses will include summaries of descriptive and aggregate antibody data against antigens from *N. gonorrhoeae* and *N. meningitidis* stratified by antigen, specimen type (serum or mucosal), pre- versus post-treatment timepoints, and treatment arm (4CMenB or placebo). No hypothesis tests

or modeling will be included in the interim immunogenicity analysis. This interim analysis of the data is not intended to impact the conduct of this trial. No statistical adjustments are planned.

As defined in the protocol, the SMC will review data at specified times during the course of the study for participant and overall study progress and will conduct ad hoc reviews as appropriate when a halting rule is met or for immediate concerns regarding observations during this study.

# 6.7. Multiple Comparisons/Multiplicity

There is only one primary endpoint at 5 timepoints. No formal hypothesis test of the primary outcome will be performed. No adjustments for multiple comparison are planned. No adjustment to the alpha level for CIs will be performed.

#### 7. STUDY PARTICIPANTS

# 7.1. Disposition of Participants

The disposition of participants in the study will be tabulated by Treatment group (**Table 6**). The table shows the total number of participants who screened, enrolled, received at least one dose, discontinued dosing or terminated from study follow-up, and those completing the study. The composition of analysis populations, including reasons for participant exclusion, by treatment arm, is presented in **Table 7** and **Table 8**. Participants excluded from analysis populations will also be summarized in **Listing 5**. **Table 9** shows the dates of first treatment received by group. **Table 10** will present a summary of the reasons that participants were screened but not enrolled. A listing of all participants that received study product is provided in **Listing 1**. A flowchart showing the disposition of study participants, adapted from the Consort Statement will be included (**Figure 1**). This figure will present the number of participants screened, enrolled, lost to follow-up, and analyzed, by treatment arm. A listing of participants who discontinued dosing or early terminated from study follow-up and the reason will be included in **Listing 2**. Participants who terminated early or discontinued vaccinations due to the Covid-19 pandemic will be highlighted in the listing.

#### 7.2. Protocol Deviations

A summary of participant-specific protocol deviations will be presented by the deviation category, deviation type, and Treatment group for all participants (**Table 3**). Major deviations will be reviewed for possible participant exclusion from the per protocol population, including deviations affecting eligibility at baseline, product administration deviations, primary endpoint missing data, and deviations relating to prohibited medications. See **Section 6.3.2** for per protocol exclusion definitions. All participant-specific protocol deviations and non-participant specific protocol deviations will be included in **Appendix 3** as data listings (**Listing 3** and **Listing 4**, respectively). Participants who had a protocol deviation due to the Covid-19 pandemic will be highlighted in the listing.

#### 8. IMMUNOGENICITY EVALUATION

This study was not designed to test a specific null hypothesis, rather, the objective was to characterize the immune response to GC elicited by the 4CMenB vaccine as compared with the placebo (normal saline) in healthy adult participants. Immunogenicity analysis will be presented for the Immunogenicity and PP populations. Immune responses for the study vaccine (4CMenB or placebo) will be summarized at each time point presented by study arm. Descriptive summary statistics will be provided for all assays and time points. For serum and mucosal antibody (IgG, IgA) assays by ELISA, the GMT and geometric mean fold rise (GMFR) will be calculated for each time point, (Days 1, 29, 43, 57, and 181 for GMT, and Days 29, 43, 57, and 181 for GMFR) in each study arm. Point estimates and their 95% confidence intervals will be reported for each time point. The distribution of titers will also be graphically summarized using reverse cumulative frequency distributions.

# 8.1. Primary Outcome Analysis

Rectal mucosal IgG concentrations (GMT) against GC OMV antigens at days 1, 29, 43, 57, and 181 in each Treatment group are shown in **Table 14**, **Figure 2**, and **Figure 4**. The summary of GMFR from baseline are also shown in **Table 14**. The distributions of rectal mucosal IgG titers are graphically summarized using reverse cumulative frequency distributions in **Figure 36** and **Figure 37**. All results are presented in **Listing 9**. A summary of GMT and GMFR Rectal mucosal IgG by sex is shown in table **Table 15**, **Figure 3**, and **Figure 5**.

# 8.2. Secondary Outcome Analyses

Serum IgG concentrations (GMT) against GC OMV antigens at days 1, 29, 43, 57, and 181 in each Treatment group are shown in **Table 16**, **Figure 6** and **Figure 8**. The summary of GMFR is also shown in **Table 16**. The distributions of serum IgG titers are graphically summarized using reverse cumulative frequency distributions in **Figure 38** and **Figure 39**. A summary of GMT and GMFR serum IgG by sex is shown in **Table 17**, **Figure 7**, and **Figure 9**. Summaries of the ratio of serum to mucosal IgG concentration will be generated at each time point and presented in **Table 22** and **Table 23**. All results are presented in **Listing 10**.

# 8.3. Exploratory Outcome Analyses

For the exploratory outcomes, summaries of IgG antibody concentrations (GMT) at each time point and GMFR in each treatment group are shown in **Table 18**, **Table 19**, **Table 20**, and **Table 21**. Summaries of the ratio of serum to mucosal IgG GMT results will be presented in **Table 22** and **Table 23**. Summaries of pairwise ratios of mucosal IgG concentrations among anatomical sites will be generated at each time point and presented in **Table 24** and **Table 25**. Summaries of IgA antibody concentrations and serum bactericidal antibody (GMT) at each time point and GMFR for other exploratory outcomes are shown starting in **Table 26** and concluding with **Table 33**. Serum Bactericidal Antibody GMT and GMFR will be presented in **Table 34**.

Summaries of the frequency of antigen-specific immune cells will include the mean if data are reported as percentage, or geometric mean if data are reported as cell count per million cells. The corresponding 95% confidence interval as well as the median, minimum, and maximum values will be presented. Fold rise from baseline will be summarized by arithmetic, geometric mean[2] or median. The summary of frequencies will be presented starting in **Table 35** and concluding with **Table 45**. Figures depicting the GMT (IgG, IgA) or frequency (MBC, T cells) for each assay over time will be presented beginning with **Figure 10** and continuing through **Figure 39** (GMTs), and **Figure 74** to **Figure 87** (frequencies). Reverse cumulative distribution (RCD) plots will be presented with separate panels for each visit, and separate curves within each panel for

each study arm and overall. Antibody titers are shown beginning with **Figure 40** and continuing through **Figure 73**.Percent inhibition of gonococcal adhesion to human cervical cell line (ME180) by mucosal antibodies at day 43 in each treatment group will be show in **Table 46**. The results for each participant at each visit are listed in **Listing 11** through **Listing 22**.

#### 9. SAFETY EVALUATION

All summaries and analysis of safety data will be presented for the safety analysis population. Safety summaries will be presented overall and stratified by treatment group. Listings will be sorted by treatment group, participant ID, parameter (if applicable), and visit. Continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. All categorical measures will be summarized by the frequency and percentages (based on the non-missing sample size) of observed levels.

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by treatment group overall for all enrolled participants (**Table 11** and **Table 12**). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, participants may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option. Individual participant listings will be presented for all demographics (**Listing 6**). Sexual history at baseline will be presented (**Table 47** and **Table 48**). Sexual history during follow-up visits will be presented (**Table 49** and **Table 50**).

#### 9.1.1. Pre-Existing Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 21.1 or higher. Summaries of all enrolled participants' pre-existing medical conditions will be presented by treatment group (**Table 13**). Individual participant listings will be presented for all medical conditions (**Listing 7**).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications will be presented by WHO Drug Levels 1 and 2 and treatment group for participants in the safety population (Table 69). Individual participant listings will be presented for all concomitant medications (Listing 32).

# 9.2. Measurements of Treatment Compliance

The number of doses of study product administered to participants will be presented by treatment group as part of the participant disposition table (**Table 6**). **Table 9** presents the number of participants who received a first dose at each enrollment period by treatment group. A listing of treatment compliance data by participant will also be presented in **Listing 8**.

#### 9.3. Adverse Events

Unsolicited AEs and SAEs will be coded by MedDRA for preferred term (PT) and system organ class (SOC). AEs will also be graded for severity. For each AE experienced, the participant will be asked if he/she had received medical attention, defined as hospitalization, an ER visit, or an otherwise unscheduled visit to or from medical personnel for any reason. AEs characterized by such unscheduled medical care will be designated as MAAEs. Safety will be assessed by the frequency and severity of:

- Any AE related to 4CMenB immunization through the end of the study.
- Any AE related to rectal mucosal sampling procedures through the end of the study.
- Any SAEs through the end of the study

A summary of all adverse events is provided in **Table 51**. This information is also presented graphically in **Figure 88** with number and severity of AEs categorized by MedDRA System Organ Class and treatment group. A summary of those events that occurred in  $\geq 5\%$  of participants in any treatment group is provided in **Table 54**.

#### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected 30 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a severity scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fever, chills/shivering/sweating, fatigue, malaise, myalgia and arthralgia (exclusive of the injection site), headache, and nausea. Local events include pain at injection site, pruritus, erythema, ecchymosis, induration/swelling, pain, and tenderness. **Table 56** summarizes the solicited adverse event grading scale.

The proportion of participants reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any local symptom, and any symptoms. The 95% CI will be calculated using Clopper-Pearson methodology from a binomial distribution (**Table 55**).

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the safety population. The number and percentage of participants reporting each event will be summarized by the maximum severity and treatment group, separately for each vaccination and over all vaccinations. For each event the denominator is the number of participants with non-missing data for the specific event (**Table 55**).

The number of participants reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table (**Table 56**, **Table 7**, **Table 58**, and **Table 59**) and graphically in a bar chart (**Figure 89** and **Figure 90**). A comparison of the event rate for each treatment group between dose 1 and dose 2 will be presented in **Table 60**.

Solicited adverse events by participant will be presented in Listing 23 and Listing 24.

#### 9.3.2. Unsolicited Adverse Events

When calculating the incidence of unsolicited AEs (i.e., on a per participant basis), each participant will only be counted once at the highest severity and/or relationship, and any repetitions of AEs within a participant will be ignored; the denominator will be the total number of participants in the safety population. All AEs reported will be included in the summaries and analyses.

The number and percentage of participants reporting at least one unsolicited AE will be summarized by MedDRA system organ class and preferred term. Denominators for percentages are the number of participants who received the study vaccination summarized. A 95% CI will be presented for the percentage of participants reporting any unsolicited AE (serious or non-serious) for each MedDRA system organ class and preferred term. A listing of all unsolicited AEs by participant will be presented in **Listing 25**, sorted by Treatment group, participant ID, and AE Number.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, and Treatment group:

- Participant incidence and total frequency of unsolicited adverse events with 95% CI (Table 61)
- Summary of severity and relationship to study product (Table 62)

- Participant incidence and total frequency of related unsolicited adverse events over time (Days 1-7) (Table 63)
- Participant listing of death and serious adverse events (Table 52)
- Participant listing of non-serious adverse events of moderate or greater severity (Table 53)
- Bar charts of the frequency and incidence of non-serious adverse events by severity and MedDRA system organ class (Figure 91 and Figure 92)
- Bar charts of the frequency and incidence of non-serious adverse events by relationship and MedDRA system organ class (Figure 93 and Figure 94)

# 9.4. Pregnancies

For any participants in the safety population who become pregnant during the study, every attempt will be made to follow these participants to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. A listing of pregnancies and outcomes will be presented in Listing 33, Listing 34, Listing 35, Listing 36, and Listing 37.

# 9.5. Clinical Laboratory Evaluations

Clinical laboratory evaluations assessed at the screening visit will be considered as baseline. At the screening visit (visit 00A), the following clinical laboratory parameters will be evaluated: a serology screening (HIV-1/2 and RPR), GC/CT NAAT at mucosal sites (rectum, vagina and oropharyngeal), and Trichomonas NAAT for female participants. For the rectal mucosal biopsy cohort, hematology (CBC) and coagulation testing (PT/aPTT) will be measured at visit 00A and may be repeated at visit 00B. At day 29, before the second vaccination and final visit at day 181 or early termination visit, serology screening (HIV-1/2 and RPR) and GC/CT NAAT at mucosal sites will be evaluated again. The laboratory adverse event grading scale will be presented in Table 5.

RPR, HIV antibody and STI testing will be presented in **Table 64**, **Table 65**, **Table 66**, **Table 67**, and **Table 69**. A complete listing of individual laboratory results will be presented in **Listing 26** and **Listing 27**. Participants with abnormal laboratory results, grade 1 severity or higher, will be presented in **Listing 28** and **Listing 29**, for hematology and coagulation, respectively, sorted by participant ID, parameter, and study day.

# 9.6. Vital Signs

Vital signs will be assessed at screening visits (Visit 00A or, if performed, Visits 00B and/or 00C), baseline visit (Visit 1, day 1), day 29 and 43, and possibly at other visit determined by study staff. Enrolled participants with abnormal vital signs will be listed (Listing 30).

# 9.7. Physical Examinations

Physical examinations will be performed at screening visit 00A, and possibly at every visit as determined by study staff. Physical examination will include the following organs and organ systems: general appearance, head /eyes /ears /nose /throat (HEENT), neck, lungs, heart, abdomen, extremities, musculoskeletal, lymph nodes, skin, and nervous system. Genital and rectal exams will be performed at the investigator's discretion (Listing 31).

# 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification (ATC) using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-participant listing of concomitant medication use will be presented in **Listing 32**. The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and treatment group for the Safety population (**Table 69**).

# 9.9. Other Safety Measures

There are no other safety measures performed.

# 10. OTHER ANALYSES

Not applicable

#### 11. REPORTING CONVENTIONS

The mean, geometric mean, standard deviation, and other statistics will be reported to one decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as two decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but <1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to three significant figures.

# 12. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings. R studio may also be used to generate figures.

# 13. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

There are no changes in the conduct of the study. With the protocol amendment from v6.0 to v7.0, an interim immunogenicity analysis was added. A separate interim immunogenicity report will be developed for this analysis.

#### 14. **REFERENCES**

- 1. Newman L, Rowley J, Vander Hoorn S, Wijesooriya NS, Unemo M, Low N, Stevens G, Gottlieb S, Kiarie J, Temmerman M. Global Estimates of the Prevalence and Incidence of Four Curable Sexually Transmitted Infections in 2012 Based on Systematic Review and Global Reporting. PLoS One. 2015;10(12):e0143304. doi: 10.1371/journal.pone.0143304. PubMed PMID: 26646541; PMCID: PMC4672879.
- 2. Gonorrhea: Division of STD Prevention; 2018 [cited 2019 March 22]. Available from: https://www.cdc.gov/std/stats17/gonorrhea.htm.
- 3. Petousis-Harris H, Paynter J, Morgan J, Saxton P, McArdle B, Goodyear-Smith F, Black S. Effectiveness of a group B outer membrane vesicle meningococcal vaccine against gonorrhoea in New Zealand: a retrospective case-control study. Lancet. 2017;390(10102):1603-10. doi: 10.1016/S0140-6736(17)31449-6. PubMed PMID: 28705462.
- 4. Paynter J, Goodyear-Smith F, Morgan J, Saxton P, Black S, Petousis-Harris H.Effectiveness of a Group B Outer Membrane Vesicle Meningococcal Vaccine in Preventing Hospitalization from Gonorrhea in New Zealand: A Retrospective Cohort Study. Vaccines (Basel). 2019;7(1). doi: 10.3390/vaccines7010005. PubMed PMID: 30621260.
- 5. Whelan J, Klovstad H, Haugen IL, Holle MR, Storsaeter J. Ecologic Study of Meningococcal B Vaccine and Neisseria gonorrhoeae Infection, Norway. Emerg Infect Dis. 2016;22(6):1137-9. doi: 0.3201/eid2206.151093. PubMed PMID: 27191543; PMCID: PMC4880101.
- 6. Pérez O, Campo Jd, Cuello M, González E, Nuñez N, Cabrera O, Llanes R, Acevedo R, Zayas C, Balboa J, Romeu B, Baró M, Campa C, Lantero MI, Sierra G, Galindo MA, Harandi AM, Lastre M. Mucosal approaches in Neisseria vaccinology. VacciMonitor. 2009;18(2):53-5.
- 7. Holst J, Oster P, Arnold R, Tatley MV, Naess LM, Aaberge IS, Galloway Y, McNicholas A, O'Hallahan J, Rosenqvist E, Black S. Vaccines against meningococcal serogroup B disease containing outer membrane vesicles (OMV): lessons from past programs and implications for the future. Hum Vaccin Immunother. 2013;9(6):1241-53. doi: 10.4161/hv.24129. PubMed PMID: 23857274; PMCID: PMC3901813.
- 8. Martin DR, Ruijne N, McCallum L, O'Hallahan J, Oster P. The VR2 epitope on the PorA P1.7-2,4 protein is the major target for the immune response elicited by the strain-specific group B meningococcal vaccine MeNZB. Clin Vaccine Immunol. 2006;13(4):486-91. doi:10.1128/CVI.13.4.486-491.2006. PubMed PMID: 16603616; PMCID: PMC1459632.
- 9. MacNeil JR, Rubin L, Folaranmi T, Ortega-Sanchez IR, Patel M, Martin SW. Use of Serogroup B Meningococcal Vaccines in Adolescents and Young Adults: Recommendations of the Advisory Committee on Immunization Practices, 2015. MMWR Morb Mortal Wkly Rep. 2015;64(41):1171-6. doi: 10.15585/mmwr.mm6441a3. PubMed PMID: 26492381.
- 10. GSK Vaccines. Bexsero Prescribing Information. 2015.
- 11. Longtin J, Dion R, Simard M, Betala Belinga J-F, Longtin Y, Lefebvre B, Labbe A-C, Deceuninck G, De Wals P. Possible Impact of Wide-scale Vaccination Against Serogroup B Neisseria Meningitidis on Gonorrhea Incidence Rates in One Region of Quebec, Canada. IDWeek 2017; San Diego, CA. 2017.

12. Semchenko EA, Tan A, Borrow R, Seib KL. The serogroup B meningococcal vaccine Bexsero elicits antibodies to Neisseria gonorrhoeae. Clin Infect Dis. 2018. doi: 10.1093/cid/ciy1061. PubMed PMID: 30551148.
# 15. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

# **APPENDICES**

# APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Study Design |
|---|---|
| Table 2: | Schedule of Study Procedures |
| Table 3: | Distribution of Protocol Deviations by Category, Type, and Treatment Group46 |
| Table 4: | Solicited Adverse Event Grading Scale |
| Table 5: | Laboratory Adverse Event Grading Scale |
| Table 6: | Participant Disposition by Treatment Group51 |
| Table 7: | Immunogenicity and Safety Populations by Treatment Group |
| Table 8: | Per-protocol Immunogenicity Populations by Treatment Group53 |
| Table 9: | Dates of First Treatment by Treatment Group |
| Table 10: | Ineligibility Summary of Screen Failures |
| Table 11: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group All Enrolled Participants |
| Table 12: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group All Enrolled Participants |
| Table 13: | Summary of Participants with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group |
| Table 14: | Primary Outcome - Rectal Mucosal IgG GMT and GMFR Results by Analysis Population, Time Point, and Treatment Group |
| Table 15: | Rectal Mucosal IgG GMT and GMFR Results by Analysis Population, Time Point, Sex and Treatment Group |
| Table 16: | Secondary Outcome - Serum IgG against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 17: | Serum IgG against OMV antigens: GMT and GMFR Results by Analysis Population, Time Point, Sex and Treatment Group |
| Table 18: | Exploratory Outcome - Serum IgG against NHBA antigens GMT and GMFR Results by Time Point and Treatment Group |
| Table 19: | Exploratory Outcome - Rectal Mucosal IgG against NHBA: GMT and GMFR Results by Time Point and Treatment Group |
| Table 20: | Exploratory Outcome - Vaginal Mucosal IgG GMT and GMFR Results by Time Point and Treatment Group |
| Table 21: | Exploratory Outcome - Oropharyngeal Mucosal IgG GMT and GMFR Results by Time Point and Treatment Group |

# Table of Tables (continued)

| Table 22: | Summaries of the Ratio of Serum to Mucosal IgG GMT Results by Time Point and Treatment Group - Immunogenicity Population |
|---|---|
| Table 23: | Summaries of the Ratio of Serum to Mucosal IgG Concentration GMT Results by Time Point and Treatment Group - Per-Protocol Population |
| Table 24: | Summaries of Pairwise IgG Concentration Ratios Comparing Anatomical Sites GMT Results by Time Point and Treatment Group - Immunogenicity Population68 |
| Table 25: | Summaries of pairwise IgG Concentration Ratios Comparing Anatomical Sites GMT Results with 95% Confidence Intervals by Time Point and Treatment Group - Per-Protocol Population |
| Table 26: | Serum IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 27: | Serum IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 28: | Rectal Mucosal IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 29: | Rectal Mucosal IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 30: | Vaginal Mucosal IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 31: | Vaginal Mucosal IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group |
| Table 32: | Oropharyngeal Mucosal IgA against OMV antigens: GMT and GMFR Results Time Point and Treatment Group |
| Table 33: | Oropharyngeal Mucosal IgA against NHBA antigens: GMT and GMFR Results Time Point and Treatment Group |
| Table 34: | Serum Bactericidal antibody GMT and GMFR Results against N. Gonorrhoeae by Time Point and Treatment Group |
| Table 35: | Frequencies of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group |
| Table 36: | Frequencies of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group |
| Table 37: | Frequencies of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group |
| Table 38: | Frequencies of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group – Intracellular Cytokine Staining (ICS), Immunogenicity Population |

# Table of Tables (continued)

| Table 39: | Frequencies and Function of Peripheral Blood CD4+ T cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population |
|---|---|
| Table 40: | Frequencies and Function of Peripheral Blood CD8+ T cells Specific for Antigens by Time Point and Treatment Group - ICS - Immunogenicity Population |
| Table 41: | Frequencies and Function of Peripheral Blood CD8+ T cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population |
| Table 42: | Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Immunogenicity Population |
| Table 43: | Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population |
| Table 44: | Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Immunogenicity Population |
| Table 45: | Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population81 |
| Table 46: | Percent Inhibition of Gonococcal Adhesion to Human Cervical Cell Line (ME180) by Mucosal Antibodies at Day 43 |
| Table 47: | Summary of Categorical Sexual History Variables at Screening - All Enrolled Participants |
| Table 48: | Summary of Continuous Sexual History Variables at Screening - All Enrolled Participants |
| Table 49: | Summary of Categorical Sexual History Variables at Follow Up - All Enrolled Participants |
| Table 50: | Summary of Continuous Sexual History Variables at Follow Up - All Enrolled Participants |
| Table 51: | Overall Summary of Adverse Events |
| Table 52: | Listing of Serious Adverse Events– Safety Population |
| Table 53: | Listing of Non-Serious Adverse Events of Moderate or Greater Severity – Safety Population |
| Table 54: | Adverse Events Occurring in $\geq$ 5% of Participants in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population91 |
| Table 55: | Number and Percentage of Participants Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Maximum Severity, Dose, and Treatment Group – Safety Population |
| Table 56: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing - 4CMenB, Post Dose 194 |
| Table 57: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing- 4CMenB, Post Dose 296 |

# Table of Tables (continued)

| Table 58: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing- Placebo, Post Dose 196 |
|---|---|
| Table 59: | Number and Percentage of Participants Experiencing Solicited Events by Symptom,<br>Severity, and Day - Placebo, Post Dose 2 |
| Table 60: | Number and Percentage of Participants Experiencing Solicited Events for Dose 1 Compared with Dose 2 by Treatment Group |
| Table 61: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Dose Number, and Treatment Group |
| Table 62: | Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and Treatment Group |
| Table 63: | Related Unsolicited Adverse Events Within 7 Days Post Dosing by MedDRA System Organ Class and Preferred Term, Dose, and Treatment Group |
| Table 64: | Laboratory Assessment RPR Results - Safety Population |
| Table 65: | Laboratory AssessmentHIV Antibody Testing Results - Safety Population102 |
| Table 66: | Laboratory Assessment – Chlamydia NAAT Testing Results - Safety Population .103 |
| Table 67: | Laboratory Assessment – Gonorrhea NAAT Testing Results - Safety Population104 |
| Table 68: | Laboratory Assessment – Trichomonas Testing Results - Safety Population105 |
| Table 69: | Number and Percentage of Participants with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group |

### 9.1 Overall Study Design and Plan Description

**Table 1:** Study Design

| | Rectal Mucosal<br>(N= | Biopsy Cohort<br>20)* | No Rectal Mucos<br>(N= | Total | |
|---|---|---|---|---|---|
| Vaccine | Male Non-pregnant Female | | Male | Male Non-pregnant Female | |
| 4CMenB | 8 | 8 | 12 | 12 | 40 |
| Placebo | 2 | 2 | 3 | 3 | 10 |

<sup>\*</sup>As noted in the study design, this trial will enroll approximately 50 (maximum of 60 participants) - approximately 20 in Rectal Mucosal Biopsy Cohort and approximately 30 in No Rectal Mucosal Biopsy Cohort

### 9.5.1 Immunogenicity and Safety Measurements Assessed and Flow Chart

 Table 2:
 Schedule of Study Procedures

| Procedures | Screening (Visit 00A) Day -56 to -1 (-56 to -28 for biopsy cohort) | Screening (Visit 00B) Day -7 to -1 (-34 to -28 for biopsy cohort) | Baseline Rectal Mucosal<br>Biopsy Visit 00C<br>,Day -28 to -1 | Study Visit 00P (Phone visit)<br>Day -27 to -12 | Enrollment/Baseline<br>visit I,Day I | Study Visit 2 $Day \ 8 \pm I day$ | Study Visit 3 $Day 15 \pm 1 day$ | Study Visit 4<br>Day 29 ±1day | Study Visit 5<br>Day 36±1day | Study Visit 6<br>Day 43 ±3 days | Study Visit 6p<br>Day 44±1 days | Study Visit 7<br>Day 57 ±1days | Final Study visit<br>Day 18 ±7 days | Early ITermination Visit <sup>15</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | | | | | | | | | | | | | |
| Assessment of Eligibility criteria | X | X | X | | X | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| Medical history | X | X | X | | X | X | X | X | X | X | | X | X | X |
| Sexual history | X | X | X | | X | | | X | | X | | X | X | X |
| Randomization | | | | | X | | | | | | | | | |
| Concomitant medications | X | X | X | | X | X | X | X | X | X | | X | X | X |
| Review covid-19 Vaccine history | | | | | X | | | X | | | | | | |
| Vital signs | X | (X) | X | | X | (X) | (X) | X | (X) | X | | (X) | (X) | (X) |
| Physical exam | X | (X) | (X) | | (X) | (X) | (X) | (X) | (X) | (X) | | (X) | (X) | (X) |
| Administer study intervention | | | | | X | | | Xe | | | | | | |
| Pre-vaccine reactogenicity assessment | | | | | X | | | X | | | | | | |
| Post-vaccine, Observation to assess<br>Acute reaction (for ≥15 minutes) | | | | | X | | | X | | | | | | |
| Evaluation vaccine site,<br>Reactogenicity and AE/SAE after<br>≥15 minutes | | | | | X | | | X | | | | | | |
| Memory aid | | | | | X | X | | X | X | | | | | (X) |
| AE review and evaluation | | | X <sup>d</sup> | X <sup>d</sup> | X | X | X | X | X | X | (X) | X | X | X |

Table 2: Schedule of Study Procedures (continued)

| | Procedures | Screening (Visit 00A) Day -56 to -1 (-56 to -28 for biopsy cohort) | Screening (Visit 00B) Day -7 to -1 (-34 to -28 for biopsy cohort) | Baseline Rectal Mucosal<br>Biopsy Visit 00C<br>,Day -28 to -1 | Study Visit 00P (Phone visit)<br>Day -27 to -12 | ıent/Bas<br>t I,Day | Study Visit 2<br>Day 8 ±1day | Study Visit 3<br>Day 15±1day | Study Visit 4<br>Day 29 ±1day | Study Visit 5<br>Day 36 ±Iday | Study Visit 6<br>Day 43 ±3 days | Study Visit 6p<br>Day 44±1days | Study Visit 7<br>Day 57±1days | Final Study visit<br>Day 18 ±7 days | Early 1Termination Visit <sup>15</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Hematology (CBC, PT, aPTT) <sup>a</sup> | X | (X) | (X) | | | | | | | | | | | |
| | Urine pregnancy test | X | (X) | | | X | | | X | | | | | | (X) |
| ion | STI screening <sup>b</sup> | X <sup>c</sup> | | | | (X) | (X) | (X) | (X) | (X) | (X) | | (X) | X | |
| llect | Rectal mucosal biopsy <sup>a</sup> | | | X | | | | | | | Xf | | | | |
| Specimen collection | Secretion sampling<br>(Vaginal, rectal,<br>Oropharyngeal) | | | | | X | | | X | | X | | X | X | (X) |
| Sı | Blood for serum antibody assays | | | | | X | | | X | | X | | X | X | (X) |
| | Blood for systemic immunity assays | | | | | X | X | X | X | X | X | X | X | X | (X) |

<sup>&</sup>lt;sup>a</sup> Only to be performed in the rectal mucosal biopsy cohort (N=20)

**Abbreviations**: X, study procedure for all participants; (X), study procedures to be determined by study staff; CBC, complete blood count; PT, prothrombin time; aPTT, activated partial thromboplastin time; STI, sexually transmitted infection

<sup>&</sup>lt;sup>b</sup> STI screening will include GC/CT NAAT of urine, pharynx, and rectum, and RPR. HIV antibody testing will occur at Visit 00A and 08 only

<sup>&</sup>lt;sup>c</sup> Baseline STI screening in non-pregnant females will also include NAAT for Trichomonas

<sup>&</sup>lt;sup>d</sup> AE review and evaluation at Visit 00C will include only AEs from the baseline biopsy procedure

<sup>&</sup>lt;sup>e</sup> The following will be reviewed for safety prior to administering the second dose: interim medical history, concomitant medications, COVID-19 vaccination status, vital signs, and negative pregnancy test result for females of childbearing potential.

f The following will be reviewed for safety prior to the rectal mucosal biopsy procedure: interim medical history, concomitant medications, and vital signs.

#### 10.2 Protocol Deviations

Table 3: Distribution of Protocol Deviations by Category, Type, and Treatment Group

| Category | | | 4CMenB<br>(N=X) | | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| | Deviation Type | No. of<br>Part. | No. of<br>Dev. | No. of<br>Part. | No. of<br>Dev. | No. of<br>Part. | No. of<br>Dev. |
| Eligibility/enrollment | Any type | X | Х | X | Х | Х | х |
| | Did not meet inclusion criterion | X | Х | X | Х | Х | х |
| | Met exclusion criterion | x | X | X | х | х | х |
| | ICF not signed prior to study procedures | x | X | X | х | х | х |
| | Other | x | Х | х | Х | х | х |
| Treatment administration schedule | Any type | x | Х | х | Х | х | х |
| | Out of window visit | х | Х | х | Х | Х | х |
| | Missed visit/visit not conducted | x | X | X | Х | Х | х |
| | Missed treatment administration | х | Х | х | Х | Х | х |
| | Delayed treatment administration | x | Х | х | Х | х | х |
| | Other | X | Х | X | Х | Х | х |
| Follow-up visit schedule | Any type | X | Х | X | Х | Х | х |
| | Out of window visit | x | X | X | х | х | х |
| | Missed visit/visit not conducted | x | X | х | Х | х | х |
| | Other | x | X | х | Х | х | х |
| Protocol procedure/assessment | Any type | X | Х | X | Х | Х | х |
| | Incorrect version of ICF signed | X | Х | X | Х | Х | х |
| | Blood not collected | x | X | х | Х | х | х |
| | Urine not collected | X | X | х | х | х | х |
| | Stool not collected | X | X | х | х | х | х |
| | Other specimen not collected | X | Х | х | х | х | х |
| | Too few aliquots obtained | x | X | Х | Х | X | х |

Table 3: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| Category | | 4CMenB<br>(N=X) | | | cebo<br>=X) | All Participants (N=X) | |
|---|---|---|---|---|---|---|---|
| | Deviation Type | No. of<br>Part. | No. of<br>Dev. | No. of<br>Part. | No. of<br>Dev. | No. of<br>Part. | No. of<br>Dev. |
| | Specimen result not obtained | X | Х | х | X | х | Х |
| | Required procedure not conducted | X | Х | х | X | х | Х |
| | Required procedure done incorrectly | X | Х | х | X | х | Х |
| | Study product temperature excursion | X | Х | х | X | х | Х |
| | Specimen temperature excursion | X | Х | х | X | х | Х |
| | Other | X | Х | х | X | х | Х |
| Treatment administration | Any type | X | Х | х | X | х | Х |
| | Required procedure done incorrectly | X | Х | х | X | х | Х |
| | Study product temperature excursion | X | Х | х | X | х | Х |
| | Other | X | Х | X | X | х | х |
| Blinding policy/procedure | Any type | X | X | X | X | Х | X |
| | Treatment unblinded | X | Х | х | X | х | х |
| | Other | X | Х | х | x | х | х |
| Note: N = Number of participants | in each group in the safety population | | | | | | |

### 12.2.2 Displays of Adverse Events

### **Table 4:** Solicited Adverse Event Grading Scale

[Implementation Note: Extract Solicited Adverse Event Grading Scale/grading scales from protocol and include here.]

| Local (Injection Site) Reaction | n | | |
|---|---|---|---|
| | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Pain – experienced without touching the injection site (spontaneous discomfort) | Participant is aware of pain, but it does not interfere with daily activity, <b>and</b> it does not require pain medication, or it requires use of a non-narcotic pain reliever ≤24hours | Participant is aware of pain; there is interference with daily activity, <b>or</b> it requires repeated use of a non-narcotic pain reliever for >24 hours | Participant is aware of pain, <b>and</b> it prevents daily activity or requires any use of a narcotic pain reliever |
| Tenderness – hurts only when injection site is touched or the arm is moved | The area immediately surrounding the injection site hurts only when touched or with arm motion, <b>and</b> it does <b>not</b> interfere with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, <b>and</b> it interferes with daily activity | The area immediately surrounding the injection site hurts when touched or with arm motion, <b>and</b> it prevents daily activity |
| Pruritus (Itching) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis (Bruising) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Erythema (Redness) | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Induration<br>(Hardness)/Swelling | Does not interfere with daily activity | Interferes with daily activity | Prevents daily activity |
| Ecchymosis (Bruising) <sup>a</sup> | 25 mm – 50 mm | 51 mm – 100 mm | >100 mm |
| Erythema (Redness) <sup>a</sup> | 25 mm – 50 mm | 51 mm – 100 mm | >100 mm |
| Induration<br>(Hardness)/Swelling <sup>a</sup> | 25 mm – 50 mm | 51 mm – 100 mm | >100 mm |
| Participantive Systemic React | togenicity | | |
| Feverishness (Chills/Shivering/Sweating) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue (Tiredness) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Malaise (General Unwell<br>Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Myalgia (Body<br>Aches/Muscular Pain) <sup>b</sup> | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Arthralgia (Joint Pain) <sup>b</sup> | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Headache | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |
| Nausea | No interference with daily activity | Some interference with daily activity | Significant interference, prevents daily activity |

Table 4: Solicited Adverse Event Grading Scale (continued)

| Quantitative Systemic Reacto | Quantitative Systemic Reactogenicity Grading | | |
|---|---|---|---|
| | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
| Fever <sup>c</sup> – oral <sup>d,#</sup> | 38.0°C – 38.4°C<br>100.4°F – 101.1°F | 38.5°C – 38.9°C<br>101.2°F – 102.0°F | >38.9°C<br>>102.0°F |
| Pulse and Blood Pressure Gra | nding | | |
| Bradycardia - beats per minute | 50 - 54 | 45 - 49 | <45 |
| Tachycardia - beats per minute | 101 - 115 | 116 -130 | >130 |
| Hypotension (systolic) mmHg | 85 - 89 | 80 - 84 | <80 |
| Hypotension (diastolic) mmHg | 50 - 54 | 45 - 49 | <45 |
| Hypertension (diastolic) mmHg | 141 - 150 | 151 - 155 | >155 |
| Hypertension (diastolic) mmHg | 91 - 95 | 96 - 100 | >100 |

<sup>&</sup>lt;sup>a</sup> Size will also be measured in mm but will not be used as a halting criterion.

<sup>&</sup>lt;sup>b</sup> Not at injection site.

<sup>&</sup>lt;sup>c</sup> A fever can be considered not related to the vaccine if an alternative etiology can be documented.

<sup>d</sup> Participants must not eat or drink anything hot or cold, or smoke within 10 minutes prior to taking oral temperature.

<sup>#</sup> Oral temperature, pulse and blood pressure assessed on Day 1 prior to the first study vaccination will be considered as baseline.

### 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

 Table 5:
 Laboratory Adverse Event Grading Scale

| Hematology | Normal Range | Mild (Grade 1) | Moderate (Grade 2) | Severe (Grade 3) |
|---|---|---|---|---|
| WBC $10^3/\mu L$ (Low) | 3.8 - 10.8 | 2.5 - 3.7 | 1.5 – 2.4 | <1.5 |
| WBC 10 <sup>3</sup> /μL (High) | 3.8 - 10.8 | 10.9 – 15.0 | 15.1 – 20.0 | >20.0 |
| Hgb g/dL (Low) (Female) | 11.7 – 15.5 | 11.0 – 11.6 | 9.5 – 10.9 | <9.5 |
| Hgb g/dL (Low) (Male) | 13.2 – 17.1 | 12.0 – 13.1 | 10.0 – 11.9 | <10.0 |
| Platelets 10 <sup>3</sup> /µL (Low) | 140 – 400 | 125 – 139 | 100 – 124 | <100 |
| Platelets 10 <sup>3</sup> /μL (High) | 140 - 400 | 401 – 550 | 551-750 | >750 |
| PT (seconds) (increase by factor) (prothrombin time) | 9.0 – 11.5 | >1.0 – 1.1 x ULN | >1.1 – 1.2 x ULN | > 1.2 x ULN |
| aPTT (seconds) (increase by factor) (activated partial thromboplastin time) | 22.0 – 34.0 | >1.0 – 1.2 x ULN | >1.2 – 1.4 x ULN | >1.4 x ULN |

### 14.1 Description of Study Participants

### 14.1.1 Disposition of Participants

**Table 6:** Participant Disposition by Treatment Group

| | 4CMenB | | | | | | Placebo | | | | | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Participant | Rectal Biopsy<br>Cohort (N=X) | | Non- Rectal Biopsy<br>Cohort (N=X) | | All 4CMenB (N=X) | | Rectal Biopsy<br>Cohort (N=X) | | Non- Rectal Biopsy<br>Cohort (N=X) | | All Placebo (N=X) | | | |
| Disposition | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | | | | | x | |
| Enrolled/Randomized | x | 100 | х | 100 | х | 100 | x | 100 | х | 100 | x | 100 | x | 100 |
| Received Treatment | x | xx | х | xx | х | xx | x | xx | х | xx | x | xx | x | XX |
| Received All Scheduled Treatments <sup>a</sup> | x | xx | х | xx | х | xx | x | xx | х | xx | x | xx | x | XX |
| Completed Final Specimen Collections | x | xx | х | xx | х | xx | x | xx | х | xx | x | xx | x | XX |
| Completed all Follow-up (Study Day 181) a | X | xx | х | xx | х | xx | X | xx | х | xx | x | xx | X | XX |
| Completed Per Protocol <sup>b</sup> | x | xx | х | xx | х | xx | x | xx | х | xx | x | xx | x | XX |

Note: N = Number of participants enrolled in each group

<sup>&</sup>lt;sup>a</sup> Refer to Listing 16.2.1 for reasons participants discontinued or terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing 16.2.3 for reasons participants are excluded from the Analysis populations.

Table 7: Immunogenicity and Safety Populations by Treatment Group

[Implementation Note: The reasons listed here should match the SAP text that describes who will be excluded from analyses.

| | | _ | MenB<br>N=X) | | cebo<br>=X) | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| Populations | Reason Participants Excluded | n | % | n | % | n | % |
| Overall Immunogenicity population* | Any Reason | Х | XX | х | XX | х | xx |
| | Did not receive first dose | X | XX | X | XX | X | XX |
| | No Baseline Sample | X | XX | X | XX | X | XX |
| | No Baseline Result reported | X | XX | х | XX | х | xx |
| | Other | X | XX | х | XX | х | xx |
| Immunogenicity population for assays | Any Reason | X | XX | х | XX | х | xx |
| with vaginal mucosal specimen* | Did not receive first dose | Х | XX | х | XX | х | XX |
| | No Baseline Sample | Х | XX | х | XX | x | XX |
| | No Baseline Result reported | Х | XX | х | XX | x | XX |
| | Other | Х | XX | х | XX | x | XX |
| Safety Analysis population | Did not receive first study vaccination. | X | XX | X | XX | х | XX |

Notes: The population is defined at the baseline visit, the number of participants may be different at each visit time; For each specific assay, there may be missing values for certain assays.

N = Number of participants enrolled in each group

Table 8: Per-protocol Immunogenicity Populations by Treatment Group

| | | 4CM<br>(N= | | | cebo<br>=X) | All Part<br>(N= | icipants<br>=X) |
|---|---|---|---|---|---|---|---|
| Analysis Populations | Reason Participants Excluded | n | % | n | % | n | % |
| Overall Per Protocol | Any protocol deviation | X | XX | X | XX | X | XX |
| Immunogenicity Analysis Population | Deviation with Eligibility/enrollment | X | XX | X | XX | X | XX |
| | Deviation with Treatment administration schedule | X | XX | Х | XX | X | XX |
| | Deviation with Follow-up visit schedule | X | XX | X | XX | X | XX |
| | Deviation with Treatment administration | X | XX | Х | XX | X | XX |
| | Deviation with Protocol procedure/assessment | X | xx | X | xx | X | XX |
| | Deviation with Blinding policy/procedure | X | XX | Х | XX | X | XX |
| | Other | х | xx | х | xx | Х | XX |
| Per Protocol | Any protocol deviation | х | xx | х | xx | Х | XX |
| Immunogenicity Analysis Population- | Deviation with Eligibility/enrollment | х | xx | х | xx | Х | XX |
| assays with vaginal | Deviation with Treatment administration schedule | х | xx | х | xx | х | XX |
| mucosal specimen | Deviation with Follow-up visit schedule | х | xx | x | xx | х | xx |
| | Deviation with Treatment administration | х | xx | x | xx | х | xx |
| | Deviation with Protocol procedure/assessment | х | XX | х | XX | X | xx |
| | Deviation with Blinding policy/procedure | х | XX | х | XX | X | XX |
| | Other | х | xx | x | xx | X | xx |

Notes: N = Number of participants enrolled in each group
The number of participants may be different at each visit;
For each specific assay, the number of participants may be different.

Table 9: **Dates of First Treatment by Treatment Group** 

| Dates of Dosing | 4CMenB<br>(N=X) | Placebo<br>(N=X) | All Participants<br>(N=X) |
|---|---|---|---|
| Total (Entire period of enrollment) | | | |
| DDMMMYYYY-DDMMMYYYY [categorize based on length of enrollment period] | x | X | x |

Notes: The dates of dosing will be categorized by 3 month period. N = Number of participants enrolled in each group

Table 10: **Ineligibility Summary of Screen Failures** 

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | nª | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of participants failing any eligibility criterion | X | xx |
| | Any inclusion criterion | X | xx |
| | [inclusion criterion 1] | х | xx |
| | [inclusion criterion 2] | х | xx |
| Inclusion | [inclusion criterion 3] | х | xx |
| | Any exclusion criterion | х | xx |
| | [exclusion criterion 1] | х | xx |
| | [exclusion criterion 2] | х | xx |
| Exclusion | [exclusion criterion 3] | х | xx |
| Eligible but Not Enrolled | | х | xx |
| a Mana than and anitanian may be man | | • | 1 |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per participant.
<sup>b</sup> Denominator for percentages is the total number of screen failures.

## 14.1.2 Demographic Data by Study Group

Table 11: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - All Enrolled Participants

| | 4CMen | B (N=X) | Placebo | o (N=X) | All Participants (N=X) | |
|---|---|---|---|---|---|---|
| Characteristic | n | % | n | % | n | % |
| Male | X | xx | X | xx | х | XX |
| Female | | | | | | |
| Not Hispanic or Latino | X | xx | X | xx | Х | XX |
| Hispanic or Latino | | | | | | |
| Not Reported | | | | | | |
| Unknown | | | | | | |
| American Indian or Alaska Native | Х | xx | X | xx | х | XX |
| Asian | | | | | | |
| Native Hawaiian or Other Pacific Islander | | | | | | |
| Black or African American | | | | | | |
| White | | | | | | |
| Multi-Racial | | | | | | |
| Unknown | | | | | | |
| | Male Female Not Hispanic or Latino Hispanic or Latino Not Reported Unknown American Indian or Alaska Native Asian Native Hawaiian or Other Pacific Islander Black or African American White Multi-Racial | Characteristic n Male X Female Not Hispanic or Latino X Hispanic or Latino Not Reported Unknown American Indian or Alaska Native x Asian Native Hawaiian or Other Pacific Islander Black or African American White Multi-Racial | Male X xx Female Not Hispanic or Latino X xx Hispanic or Latino Not Reported Unknown American Indian or Alaska Native x xx Asian Native Hawaiian or Other Pacific Islander Black or African American White Multi-Racial | Characteristic n % n Male X xx x Female Not Hispanic or Latino X xx x Hispanic or Latino Not Reported Unknown American Indian or Alaska Native x xx x Asian Native Hawaiian or Other Pacific Islander Black or African American White Multi-Racial | Characteristic n % n % Male X XX XX XX Female Not Hispanic or Latino X XX XX XX Hispanic or Latino Not Reported Unknown American Indian or Alaska Native X XX XX XX Asian Native Hawaiian or Other Pacific Islander | Characteristic n % n % n Male X xx xx x xx xx x Female Not Hispanic or Latino X xx xx x xx x Hispanic or Latino Not Reported Unknown American Indian or Alaska Native x xx xx x xx x Asian Native Hawaiian or Other Pacific Islander Black or African American White Multi-Racial |

Table 12: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group - All Enrolled Participants

| Variable | Statistic | 4CMenB<br>(N=X) | Placebo<br>(N=X) | All Participants (N=X) |
|---|---|---|---|---|
| Age (years) | Mean | xx | xx | xx |
| | Standard Deviation | xx | xx | xx |
| | Median | х | X | х |
| | Minimum | Х | X | х |
| | Maximum | X | X | х |
| Note: N = Number of pa | articipants in each group | • | • | • |

### 14.1.3 Prior and Concurrent Medical Conditions

Table 13: Summary of Participants with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| | 4CM<br>(N= | | | cebo<br>=X) | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|
| MedDRA System Organ Class | n | % | n | % | n | % |
| Any SOC | X | XX | X | XX | X | XX |
| [SOC 1] | | | | | | |
| [SOC 2] | | | | | | |

Notes: n = Number of participants reporting medical history within the specified SOC. A participant is only counted once per SOC. <math>N = Total number of participants in each group.

Table 14: Primary Outcome - Rectal Mucosal IgG GMT and GMFR Results by Analysis Population, Time Point, and Treatment Group

| | | | 4CM | enB | Pla | acebo |
|---|---|---|---|---|---|---|
| Population | <b>Time Point</b> | Statistic | OMV Ng 1291 | OMV Ng CNG20 | OMV Ng 1291 | OMV Ng CNG20 |
| nmunogenicity Population | Day 1 | N | X | X | X | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) |
| | <b>Day 29</b> | N | X | X | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | X | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| er-Protocol Population | Day 1 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | X | X | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | X | X | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Note: N = Number of participants in the Immunogenicity Population for Rectal Mucosal data for a specific assay (OMV1291, and OMV20) at each time for certain Treatment Group

**Table 15:** Rectal Mucosal IgG GMT and GMFR Results by Analysis Population, Time Point, Sex and Treatment Group

| | | | | 4CM | enB | | | Placel | 00 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Fen | ıale | N | <b>Tale</b> | Fe | male | N | <b>Tale</b> |
| Population | Time Point | Statistic | OMV 1291 | OMV CNG20 | OMV 1291 | OMV CNG20 | OMV 1291 | OMV CNG20 | OMV 1291 | OMV CNG20 |
| Immunogenicity | Day 1 | N | x | х | X | х | X | х | х | х |
| Population | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | X | х | х | х | X | х | Х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | х | х | х | X | х | Х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | х | х | х | X | х | Х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | х | X | х | X | х | х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| Per-Protocol | Day 1 | N | х | х | х | х | X | х | Х | х |
| Population | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | X | x | X | X | X | X | X | X |
| | | GMT (95% CI) | x (x, x) | x(x, x) | x(x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | х | X | X | X | x | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | x | X | X | X | X | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | x | х | х | х | X | х | х | х |
| Day 18 | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Table 16: Secondary Outcome - Serum IgG against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group

| | | | | 4CMenB | | | Placebo | |
|---|---|---|---|---|---|---|---|---|
| Population | Time Point | Statistic | OMV NZ98 | OMV Ng 1291 | OMV Ng CNG20 | OMV NZ98 | OMV Ng 1291 | OMV Ng CNG20 |
| Immunogenicity | Day 1 | N | Х | х | х | Х | Х | X |
| Population | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | <b>Day 29</b> | N | X | X | x | X | Х | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | Day 43 | N | X | X | x | X | X | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | Day 57 | N | X | x | x | X | X | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | Day 181 | N | X | x | x | X | X | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| Per-Protocol | Day 1 | N | X | x | x | X | X | X |
| Population | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) |
| | <b>Day 29</b> | N | X | X | x | X | Х | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | x | x | X | X | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) |
| | Day 57 | N | Х | X | x | X | Х | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | х | х | х | х | х | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Note: N = Number of participants in the Immunogenicity Population for Rectal Mucosal data for a specific assay (OMV98, OMV1291, and OMV20) at each time for certain Treatment Group

Table 17: Serum IgG against OMV antigens: GMT and GMFR Results by Analysis Population, Time Point, Sex and Treatment Group

| | | | | | 4CMe | nB | | | | | Place | bo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | İ | | Female | | | Male | | | Female | | | Male | |
| Population | Time<br>Point | Statistic | OMV NZ98 | OMV 1291 | OMV CNG20 | OMV<br>NZ98 | OMV 1291 | OMV CNG20 | OMV<br>NZ98 | OMV 1291 | OMV CNG20 | OMV<br>NZ98 | OMV 1291 | OMV CNG20 |
| Immunogenicity | Day 1 | N | X | X | X | X | Х | X | X | X | x | X | Х | х |
| Population | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x (x, x) | x(x, x) |
| | Day 29 | N | X | X | X | X | х | X | X | x | х | х | х | х |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | X | х | X | х | х | X | X | х | X | Х | х |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | X | х | х | Х | х | X | X | х | х | х | х |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | X | х | X | Х | х | X | X | х | Х | х | х |
| D | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Serum IgG against OMV antigens: GMT and GMFR Results by Analysis Population, Time Point, Sex and Treatment Group (continued) Table 17:

| | | | | | 4CM | enB | | | | | Plac | ebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Per-Protocol<br>Population | Day 1 | N | X | X | х | X | X | X | X | X | X | X | X | X |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | Х | X | х | Х | X | X | Х | X | Х | х | Х | Х |
| | | GMT (95%<br>CI) | x(x, x) | x (x, x) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | Х | X | х | х | Х | X | X | X | X | х | Х | Х |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | Х | X | х | х | Х | X | X | X | X | х | Х | X |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | Х | X | х | х | X | X | X | X | X | х | X | X |
| | | GMT (95%<br>CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR<br>(95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Table 18: Exploratory Outcome - Serum IgG against NHBA antigens GMT and GMFR Results by Time Point and Treatment Group

| | | | | 4CMenB | | | Placebo | |
|---|---|---|---|---|---|---|---|---|
| Population | Time Point | Statistic | NHBA NZ98 | NHBA Ng 1291 | NHBA Ng CNG20 | NHBA NZ98 | NHBA Ng 1291 | NHBA Ng CNG20 |
| Immunogenicity | Day 1 | N | х | х | х | Х | х | х |
| Population | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | <b>Day 29</b> | N | х | X | х | Х | х | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | X | X | X | X | X |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) |
| | Day 57 | N | X | X | X | X | X | х |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | X | X | X | X | х |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| Per-Protocol | Day 1 | N | X | X | X | X | X | X |
| Population | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x(x, x) | x(x, x) |
| | <b>Day 29</b> | N | X | X | х | X | Х | Х |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | X | X | X | X | х |
| | | GMT (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x(x, x) | x (x, x) | x (x, x) | x(x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | х | X | х | X | Х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | х | х | х | Х | х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Note: N = Number of participants in the Immunogenicity Population for Rectal Mucosal data for a specific assay (NHBA NZ98, NHBA Ng1291, and NHBA CNG20) at each time for certain Treatment Group

Note: Following tables have the similar format with Table 14

#### Table 19: Exploratory Outcome - Rectal Mucosal IgG against NHBA: GMT and GMFR Results by Time Point and Treatment Group

[note: The assays may be performed depending on specimen availability and interim immunogenicity analysis report]

#### Table 20: Exploratory Outcome - Vaginal Mucosal IgG GMT and GMFR Results by Time Point and Treatment Group

[note: Vaginal mucosal include lavage and swab samples, this table will summarize the two types of samples in separated rows; if only one type of sample is tested, then only that type will be included.

The assays for IgG against OMV antigen will be performed, the assay against NHBA antigen maybe performed depending on specimen availability and interim immunogenicity analysis report]

### Table 21: Exploratory Outcome - Oropharyngeal Mucosal IgG GMT and GMFR Results by Time Point and Treatment Group

[note: The assays for IgG against OMV antigen will be performed, the assay against NHBA antigen maybe performed depending on specimen availability and interim immunogenicity analysis report]

Table 22: Summaries of the Ratio of Serum to Mucosal IgG GMT Results by Time Point and Treatment Group - Immunogenicity Population

| | | | | 4CMenB | | Placebo | | |
|---|---|---|---|---|---|---|---|---|
| Assay | Time | Statistic | Serum vs Rectal<br>Mucosal IgG | Serum vs<br>Oropharyngeal IgG | Serum vs Vaginal<br>Mucosal IgG | Serum vs Rectal<br>Mucosal IgG | Serum vs<br>Oropharyngeal IgG | Serum vs Vaginal<br>Mucosal IgG |
| OMV Ng1291 | Day 1 | N | Х | х | X | х | x | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | X | X | Х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| OMV Ng | Day 1 | N | X | X | X | Х | X | х |
| CNG20 | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | X | х | X | Х | х | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | X | х | X | Х | x | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Note: N = Number of participants in the Immunogenicity Population for specific pair of immunoassays, when comparing serum vs rectal and oropharyngeal mucosal, both male and female are included, when compare with Vaginal mucosal IgG, only females are included.

Same format for following table:

Table 23: Summaries of the Ratio of Serum to Mucosal IgG Concentration GMT Results by Time Point and Treatment Group - Per-Protocol Population

Table 24: Summaries of Pairwise IgG Concentration Ratios Comparing Anatomical Sites GMT Results by Time Point and Treatment Group - Immunogenicity Population

| | | | | 4CMenB | | Placebo | | |
|---|---|---|---|---|---|---|---|---|
| Assay | Time | Statistic | Rectal vs<br>Oropharyngeal IgG | Rectal vs Vaginal<br>Mucosal IgG | Vaginal vs<br>Oropharyngeal IgG | Rectal vs<br>Oropharyngeal IgG | Rectal vs Vaginal<br>Mucosal IgG | Vaginal vs<br>Oropharyngeal IgG |
| OMV<br>Ng1291 | Day 1 | N | х | X | х | Х | X | х |
| Ng1291 | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | х | X | х | х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| I | Day 43 | N | х | X | х | х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | х | X | x | х | X | x |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day | N | х | X | х | х | X | х |
| | 181 | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| OMV20 | Day 1 | N | х | X | х | х | X | х |
| Ng CNG20 | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | <b>Day 29</b> | N | х | X | х | х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | х | X | х | х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | х | X | x | х | X | х |
| | | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day | N | х | X | х | х | X | х |
| OMV20<br>Ng CNG20 | 181 | Geometric Mean Ratio (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Note: N = Number of participants in the Immunogenicity Population for specific pair of immunoassays, when comparing rectal and oropharyngeal sites, both males and females are included; when comparing with vaginal site, only females are included.

Same format for following table:

Table 25: Summaries of pairwise IgG Concentration Ratios Comparing Anatomical Sites GMT Results with 95% Confidence Intervals by Time Point and Treatment Group - Per-Protocol Population

Table 26: Serum IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group

| | | | 4C | MenB | PI | acebo |
|---|---|---|---|---|---|---|
| Population | Time | Statistic | OMV Ng 1291 | OMV Ng CNG20 | OMV Ng 1291 | OMV Ng CNG20 |
| Immunogenicity | Day 1 | N | х | х | X | X |
| Population | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | OMV Ng CNG20 OMV Ng 1291 x x x (x, x) x (x, x) | x (x, x) | |
| | | GMFR (95% CI) | x (x, x)<br>x | x (x, x) | x (x, x) | x (x, x) |
| | Day 43 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 181 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| Per-Protocol Population | Day 1 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 29 | N | х | х | x | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x x x | x (x, x) | |
| | Day 43 | N | х | х | х | х |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | Day 57 | N | х | X | X | x |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Table 26: Serum IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group (continued)

| | | | 4CN | <b>I</b> enB | Placebo | |
|---|---|---|---|---|---|---|
| Population | Time | Statistic | OMV Ng 1291 | OMV Ng CNG20 | OMV Ng 1291 | OMV Ng CNG20 |
| | Day 181 | N | X | X | х | X |
| | | GMT (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| | | GMFR (95% CI) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| Note: N = Number of particit | pants in the Immunogenicity | Population for Rectal Mucosal data | for a specific assay (OMV) | 08. OMV1291, and OMV20) | for certain Treatment Gro | oun |

Same format for the following tables:

- Table 27: Serum IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group
- Table 28: Rectal Mucosal IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group
- Table 29: Rectal Mucosal IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group

[note: The assays may be performed depending on specimen availability and interim immunogenicity analysis report]

- Table 30: Vaginal Mucosal IgA against OMV antigens: GMT and GMFR Results by Time Point and Treatment Group
- Table 31: Vaginal Mucosal IgA against NHBA antigens: GMT and GMFR Results by Time Point and Treatment Group

[note: The assays may be performed depending on specimen availability and interim immunogenicity analysis report]

- Table 32: Oropharyngeal Mucosal IgA against OMV antigens: GMT and GMFR Results Time Point and Treatment Group
- Table 33: Oropharyngeal Mucosal IgA against NHBA antigens: GMT and GMFR Results Time Point and Treatment Group

[note: The assays may be performed depending on specimen availability and interim immunogenicity analysis report]

Table 34: Serum Bactericidal antibody GMT and GMFR Results against N. Gonorrhoeae by Time Point and Treatment Group

Table 35: Frequencies of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group

| | Assay: | | | 4CMen | B | Placebo | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Population | IgG MBC<br>ELISpot | Statistic | Day 1 | Day 29 | Day 43 | Day 181 | Day 1 | Day 29 | Day 43 | Day 181 |
| Immunogenicity | OMV NZ98 | N | х | x | Х | Х | Х | Х | х | Х |
| Population | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | OMV Ng1291 | N | х | x | Х | Х | Х | Х | х | Х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | OMV CNG20 | N | х | х | Х | Х | х | Х | X | Х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | NHBA NZ98 | N | х | x | х | X | X | Х | X | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | NHBA Ng1291 | N | x | x | х | X | X | х | X | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | NHBA CNG20 | N | x | X | х | X | X | х | X | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
Table 35: Frequencies of Memory B Cells Specific for OMV and NHBA antigens by Time Point and Treatment Group (continued)

| | Assay: | | | 4CMen | В | | | Placel | bo | |
|---|---|---|---|---|---|---|---|---|---|---|
| Population | IgG MBC<br>ELISpot | Statistic | Day 1 | Day 29 | Day 43 | Day 181 | Day 1 | Day 29 | Day 43 | Day 181 |
| Per-protocol | OMV NZ98 | N | x | x | Х | Х | X | x | X | X |
| Population | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | OMV Ng1291 | N | х | х | х | Х | х | Х | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | OMV CNG20 | N | х | х | х | Х | х | Х | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) x(x) x | | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | NHBA NZ98 | N | х | х | х | Х | х | Х | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) $x(x, x)$ | | x(x, x) | x(x, x) |
| | NHBA Ng1291 | N | х | х | х | Х | х | Х | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | NHBA CNG20 | N | х | х | х | X | X | х | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (Range) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |

Notes: N is the number of participants in each group at given timepoint.

Table 36: Frequencies of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group

| | Assay: | | | | | 4CMenB | | | | | | | Placebo | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Population | IFNg<br>ELISpot | Statistic | Day 1 | Day 8 | Day 15 | Day 29 | Day 36 | Day 43 | Day 57 | Day 1 | Day 8 | Day 15 | Day 29 | Day 36 | Day 43 | Day 57 |
| Immunogenicity | IFNg | N | X | X | X | х | х | Х | X | X | X | X | Х | X | X | х |
| Population | NZ98<br>OMV | Geometric Mean | х | x | х | х | х | х | х | x | х | X | х | х | х | х |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNg | N | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| | Ng1291<br>OMV | Geometric Mean | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| | ONIV | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNg | N | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| | CNG20<br>OMV | Geometric Mean | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| Per-protocol | IFNg | N | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| Population | NZ98<br>OMV | Geometric Mean | х | x | х | х | х | х | х | x | х | X | х | х | х | х |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNg | N | х | х | х | х | х | х | х | X | х | x | х | х | х | х |
| | Ng1291<br>OMV | Geometric Mean | x | x | x | х | x | x | х | x | х | x | x | x | x | х |
| | OMV | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNg | N | X | X | x | x | X | X | x | X | х | x | x | X | X | Х |
| | CNG20<br>OMV | Geometric Mean | X | X | x | x | X | X | x | X | х | x | x | X | X | Х |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |

Note: N is the number of participant in each treatment group at certain timpoint The frequencies are measured as Spots per million PBMC, format is 0 - xxxx

Table 37: Frequencies of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group

| | | | | 4CMenB | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|---|
| Population | Assay:<br>IFNg ELISpot | Statistic | Day 1 | Day 15 | Day43 | Day 1 | Day 15 | Day43 | |
| mmunogenicity | NZ98 NHBA | N | x | x | x | X | x | X | |
| Population | Peptide pool | Geometric Mean | x | х | x | х | х | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | 1291 NHBA | N | X | X | X | х | X | X | |
| | Peptide pool | Geometric Mean | х | х | х | х | х | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | CNG20 NHBA | N | x | х | х | х | х | x | |
| | Peptide pool | Geometric Mean | х | х | х | х | х | х | |
| er-Protocol | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | <b>Consensus Peptide</b> | N | х | х | х | Х | х | x | |
| | pool | Geometric Mean | х | х | х | х | х | х | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | NZ98 NHBA | N | x | Х | Х | x | X | X | x |
| <b>Population</b> | Peptide pool | Geometric Mean | x | x | x | X | X | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | 1291 NHBA | N | х | х | х | Х | х | x | |
| | Peptide pool | Geometric Mean | x | x | x | X | X | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | CNG20 NHBA | N | X | x | X | X | X | x | |
| | Peptide pool | Geometric Mean | x | x | x | X | X | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |
| | Consensus Peptide | N | x | X | X | x | X | X | |
| | pool | Geometric Mean | X | X | X | x | X | x | |
| | | 95% CI | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | |

Table 38: Frequencies of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group – Intracellular Cytokine Staining (ICS), Immunogenicity Population

| | | | | | 4CMenB | | | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assay:<br>ICS | Phenotype | Statistic | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 |
| NZ98 OMV | IL17+ as a % of CD4+ | N | х | х | х | х | х | х | x | х | х | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | TNFa+ as a % of CD4+ | N | х | х | х | х | х | х | x | X | х | x |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | IFNG+ as a % of CD4+ | N | х | х | х | х | х | х | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| 1291 OMV | IL17+ as a % of CD4+ | N | х | х | х | х | х | х | x | X | х | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | TNFa+ as a % of CD4+ | N | х | х | х | х | х | х | x | X | х | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | IFNG+ as a % of CD4+ | N | X | X | X | X | X | x | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| CNG20 OMV | IL17+ as a % of CD4+ | N | X | X | X | X | X | x | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | TNFa+ as a % of CD4+ | N | x | Х | X | х | Х | X | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | IFNG+ as a % of CD4+ | N | х | Х | х | x | х | х | X | х | X | X |

Table 38: Frequencies of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens from GC by Time Point and Treatment Group – Intracellular Cytokine Staining (ICS), Immunogenicity Population (continued)

| | | | | | 4CMenB | | | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assay:<br>ICS | Phenotype | Statistic | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| NHBA NZ98 | IL17+ as a % of CD4+ | N | X | х | х | х | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | х | х | х | X | х | х | X | х | х | x |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | X | х | х | х | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) (x, x) | | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| NHBA Ng1291 | IL17+ as a % of CD4+ | N | X | х | х | X | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | X | х | х | х | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | X | х | х | х | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| NHBA CNG20 | IL17+ as a % of CD4+ | N | X | х | х | X | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | х | х | х | х | х | х | X | х | х | х |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |

Table 38: Frequencies of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens from GC by Time Point and Treatment Group – Intracellular Cytokine Staining (ICS), Immunogenicity Population (continued)

| | | | | | 4CMenB | | | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assay:<br>ICS | Phenotype | Statistic | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 | Day 1 | Day 15 | Day 29 | Day 43 | Day 57 |
| | IFNG+ as a % of CD4+ | N | х | х | X | x | x | X | X | х | х | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| Consensus | IL17+ as a % of CD4+ | N | Х | x | X | X | X | X | X | X | X | X |
| peptide pool | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | Х | x | X | X | X | X | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | Х | x | X | X | X | X | X | X | X | X |
| | | Mean (SD) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) | x(x) |
| | | Median (IQR) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) | (x, x) |
| Note: Frequencies are | presented as percentage form | nat 0.00% - 99.99% | | | | | | | | | | |

[Implementation note for above and below table, the values reported in the table are values derived from (original value - background value)]
Same format for the following tables:

- Table 39: Frequencies and Function of Peripheral Blood CD4+ T cells Specific for Antigens by Time Point and Treatment Group ICS Per-Protocol Population
- Table 40: Frequencies and Function of Peripheral Blood CD8+ T cells Specific for Antigens by Time Point and Treatment Group ICS Immunogenicity Population

[note: The CD8 table should not contain IL17+ as cytokine]

Table 41: Frequencies and Function of Peripheral Blood CD8+ T cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population

[note: The CD8 table should not contain IL17+ as cytokine]

Table 42: Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Immunogenicity Population

[Implementation note, the values reported in the table are values derived from (original value - background value)

The assays may be performed depending on specimen availability and interim immunogenicity analysis report]

| | | | 4CN | <b>1</b> enB | Pla | icebo |
|---|---|---|---|---|---|---|
| Assay:<br>Intracellular cytokine staining (ICS) | Phenotype | Statistic | Day 1 | Day 43 | Day 1 | Day 43 |
| OMV Ng1291 | IL17+ as a % of CD4+ | N | х | х | x | х |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | x | x | x | X |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | x | x | x | X |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| OMV CNG20 | IL17+ as a % of CD4+ | N | x | X | X | X |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | x | X | x | X |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | х | x | x | х |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |

Table 42: Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Immunogenicity Population (continued)

| | | | 4CM | <b>IenB</b> | Pla | cebo |
|---|---|---|---|---|---|---|
| Assay:<br>Intracellular cytokine staining (ICS) | Phenotype | Statistic | Day 1 | Day 43 | Day 1 | Day 43 |
| NHBA Ng1291* peptide | IL17+ as a % of CD4+ | N | X | x | X | x |
| · 1 1 | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | X | х | x | х |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | X | х | x | x |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| NHBA CNG20* peptide | IL17+ as a % of CD4+ | N | X | x | X | x |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | TNFa+ as a % of CD4+ | N | X | x | X | x |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |
| | IFNG+ as a % of CD4+ | N | X | x | X | X |
| | | Median (IQR) | x(x, x) | x(x, x) | x(x, x) | x(x, x) |
| | | Range | (x, x) | (x, x) | (x, x) | (x, x) |

Same format for the following tables:

- Table 43: Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for Antigens by Time Point and Treatment Group ICS Per-Protocol Population
- Table 44: Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for Antigens by Time Point and Treatment Group ICS Immunogenicity Population

[note: The CD8 table should not contain IL17+ as cytokine]

Table 45: Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for Antigens by Time Point and Treatment Group - ICS - Per-Protocol Population

[note: The CD8 table should not contain IL17+ as cytokine]

Table 46: Percent Inhibition of Gonococcal Adhesion to Human Cervical Cell Line (ME180) by Mucosal Antibodies at Day 43

| Population | Assay | Percent Inhib | oition (95% CI) |
|---|---|---|---|
| | | 4CMenB | Placebo |
| Immunogenicity | ACMenB | | X |
| Population | BAA_1291 | x(x , x) | x(x , x) |
| | BAA_20 | x(x, x) | x(x, x) |
| Per-Protocol | N* | Х | x |
| Population | BAA_1291 | x(x , x) | x(x , x) |
| | BAA_20 | x(x , x) | x(x , x) |
| *N =Number of par | ticipants in the certain | Freatment Group for certain analysis popu | ılation |

Table 47: Summary of Categorical Sexual History Variables at Screening - All Enrolled Participants

| | | | 4CM<br>N= | | Plac<br>N= | | All Par | ticipants |
|---|---|---|---|---|---|---|---|---|
| | Variable | Characteristic | n | % | n | % | n | % |
| | Yes/No | No | X | X | X | Х | x | X |
| | i es/ino | Yes | X | X | X | X | x | X |
| Oral receptive | How often did the participant or | Always | Х | Х | Х | х | x | X |
| | the participant's partner use a condom or barrier for protection? | Sometimes | Х | Х | Х | х | x | X |
| | • | Never | х | х | х | х | х | х |
| | V AI | No | Х | Х | Х | х | x | х |
| | Yes/No | Yes | X | х | х | х | x | х |
| Oral active | How often did the participant or | Always | X | х | х | х | x | х |
| | the participant's partner use a condom or barrier for protection? | Sometimes | X | х | х | х | x | х |
| | 1 | Never | X | х | х | х | x | х |
| | V AI | No | X | х | х | х | x | х |
| | Yes/No | Yes | Х | х | х | х | x | х |
| Rectal receptive | How often did the participant or | Always | X | х | х | Х | х | х |
| тесерите | the participant's partner use a condom or barrier for protection? | Sometimes | X | х | х | х | x | х |
| | 1 | Never | x | х | х | х | х | х |
| | V. Al | No | X | х | х | х | x | х |
| | Yes/No | Yes | Х | Х | Х | х | x | х |
| Rectal insertive | How often did the participant or | Always | X | х | х | х | x | х |
| insertive | the participant's partner use a condom or barrier for protection? | Sometimes | X | х | х | х | x | х |
| | 1 | Never | X | х | х | X | х | х |
| | V /N - | No | Х | х | х | х | x | х |
| | Yes/No | Yes | х | х | х | х | х | х |
| Genital/<br>vaginal | How often did the participant or | Always | х | х | х | х | х | х |
| , 4511141 | the participant's partner use a condom or barrier for protection? | Sometimes | X | X | X | х | х | X |
| | 101 protection: | Never | X | X | X | х | x | X |
| Note: N is | the number of participants answ | ered "Yes" to the q | uestion "Sex | ual intercou | rse in last 6 | months?" | | |

Table 48: Summary of Continuous Sexual History Variables at Screening - All Enrolled Participants

| Variable | Statistics | 4CMenB<br>(N=x) | Placebo<br>(N=x) | All Participants (N=x) |
|---|---|---|---|---|
| How many total sexual partners has the participant had in the | Mean (SD) | x(x) | x(x) | x(x) |
| preceding 6 months? | Median (min, max) | x(x,x) | x(x,x) | x(x,x) |

**Table 49:** Summary of Categorical Sexual History Variables at Follow Up - All Enrolled Participants

| | | | | | Vis | it 01 | | | | | Visi | t 04 | | | | | Vis | sit 04Z | Z | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Variable | Characteristic | 4CM | enB | Plac | cebo | | All<br>cipants | 4CN | IenB | Place | ebo | | All<br>icipants | 4CI | MenB | Pla | cebo | A<br>Partic | ll<br>ipants |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sexual intercourse <sup>a,c</sup> | | Yes | x | Х | х | X | X | х | X | X | X | X | х | X | X | X | X | X | х | X |
| New partner | | Opposite-sex | X | X | X | X | X | X | X | X | X | X | Х | X | X | X | X | X | X | X |
| sexual | | Same-sex | X | Х | Х | X | X | X | X | X | X | х | Х | X | X | X | X | Х | X | х |
| orientation <sup>b</sup> | | Both | X | X | X | X | X | X | X | X | X | X | X | X | X | x | X | X | X | x |
| | Yes/No | No | X | X | X | X | х | X | X | X | X | X | X | X | X | x | X | X | x | x |
| | 1 CS/NO | Yes | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | x |
| Oral receptive | How often did the participant or the | Always | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| | participant's partner use a condom or barrier for protection? | Sometimes | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| | or barrier for protection? | Never | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| | Yes/No | No | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| | i es/No | Yes | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| Oral active | How often did the participant or the | Always | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X | X | X |
| | participant's partner use a condom or barrier for protection? | Sometimes | X | Х | Х | X | х | X | Х | X | X | х | х | X | X | X | X | Х | X | х |
| | • | Never | X | Х | Х | X | х | X | Х | X | X | х | х | X | X | X | X | Х | X | х |
| | Yes/No | No | X | Х | Х | X | х | X | Х | X | X | х | х | X | X | X | X | Х | X | х |
| | 1 es/No | Yes | X | х | х | X | х | X | Х | X | X | х | Х | X | Х | X | X | х | X | х |
| | Engage in receptive anal <= 1 week | No | X | х | Х | X | х | X | х | X | X | X | х | X | х | X | X | х | X | х |
| Rectal receptive | after the rectal biopsy procedure? How often did the participant or the | Yes | Х | х | Х | Х | х | X | Х | Х | X | х | х | X | х | х | x | х | х | х |
| | | Always | х | х | Х | х | х | х | Х | Х | X | х | х | х | х | х | x | х | х | x |
| | participant's partner use a condom or barrier for protection? | Sometimes | х | х | Х | х | х | х | Х | Х | X | х | х | х | х | х | x | х | х | x |
| | 1 | Never | X | х | Х | Х | х | X | х | X | X | Х | х | X | х | X | X | х | х | х |

Table 49: Summary of Categorical Sexual History Variables at Follow Up - All Enrolled Participants (continued)

| | | | | | Vis | it 01 | | | | | Visi | t 04 | | | | | Vis | sit 04Z | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Variable | Characteristic | 4CM | enB | Pla | cebo | | All<br>cipants | 4CM | IenB | Place | ebo | | All<br>icipants | 4CI | MenB | Pla | cebo | A<br>Partic | All<br>cipants |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Yes/No | No | Х | X | X | X | X | X | x | X | X | х | X | X | X | X | X | X | X | X |
| | Y es/No | Yes | х | X | х | X | x | х | х | x | X | х | X | X | х | х | X | X | х | X |
| Rectal insertive | How often did the participant or the | Always | х | х | Х | Х | х | х | х | х | X | X | Х | х | х | х | X | X | х | X |
| | participant's partner use a condom or barrier for protection? | Sometimes | х | X | Х | X | х | х | х | х | Х | х | Х | Х | Х | х | X | X | х | х |
| | • | Never | х | X | Х | X | х | х | х | х | Х | х | Х | Х | Х | х | X | X | х | х |
| | 37 (31 | No | х | Х | х | Х | x | Х | х | х | X | х | х | х | х | х | х | X | х | х |
| | Yes/No | Yes | х | Х | х | Х | x | Х | х | х | X | х | х | х | х | х | х | X | х | х |
| Genital/vaginal | How often did the participant or the | Always | х | X | Х | Х | х | Х | х | х | X | х | х | х | х | Х | х | X | Х | X |
| | participant's partner use a condom or barrier for protection? | Sometimes | х | Х | х | Х | х | х | х | X | Х | х | х | х | х | х | х | X | х | х |
| | • | Never | Х | х | х | X | X | х | Х | X | X | х | х | X | х | X | х | X | х | X |

<sup>&</sup>lt;sup>a</sup> The question is: Sexual intercourse since previous visit?

<sup>&</sup>lt;sup>b</sup> The question is:if there is new partner since previous visit, what is sexual orientation?

c if the answer to this question is "Yes" then continue.

**Table 50:** Summary of Continuous Sexual History Variables at Follow Up - All Enrolled Participants

| | | | Visit 01 | | | Visit 04 | | | Visit 04Z | |
|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Statistics | 4CMenB<br>(N=x) | Placebo<br>(N=x) | All<br>Participants<br>(N=x) | 4CMenB<br>(N=x) | Placebo<br>(N=x) | All<br>Participants<br>(N=x) | 4CMenB<br>(N=x) | Placebo<br>(N=x) | All<br>Participants<br>(N=x) |
| How many total sexual partners has the | Mean (SD) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) |
| participant had since previous visit? | Median (min, max) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) |
| How many new sexual partners has the | Mean (SD) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x (x) | x(x) |
| participant had? * | Median (min, max) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) | x (x,x) |

<sup>\*</sup> New partner defined as partners since the last assessment with no sexual contact in the 6 months prior to initial screening.

## 14.3 Safety Data

## 14.3.1 Displays of Adverse Events

**Table 51:** Overall Summary of Adverse Events

| | _ | MenB<br>= x) | | cebo<br>= x) | | ticipants<br>= x) |
|---|---|---|---|---|---|---|
| Participants <sup>a</sup> with | n | % | n | % | n | % |
| At least one solicited adverse event | | | | | | |
| At least one local solicited adverse event | x | х | х | х | х | х |
| At least one systemic solicited adverse event | x | х | х | х | х | Х |
| At least one solicited adverse event due to rectal mucosal biopsy procedure | х | х | х | х | х | Х |
| At least one unsolicited adverse event | x | х | х | х | х | х |
| Mild (Grade 1) | x | х | х | х | х | х |
| Moderate (Grade 2) | x | х | х | х | х | Х |
| Severe (Grade 3) | x | х | х | х | х | Х |
| Not yet assessed | X | х | х | х | х | Х |
| At least one related unsolicited adverse event | X | х | х | х | х | Х |
| Mild (Grade 1) | x | х | х | х | х | Х |
| Moderate (Grade 2) | X | Х | х | X | x | Х |
| Severe (Grade 3) | X | х | х | х | х | Х |
| Not yet assessed | X | Х | х | X | x | Х |
| At least one severe (Grade 3) unsolicited adverse event | X | х | х | х | х | Х |
| Related | X | х | х | х | х | Х |
| Unrelated | X | х | х | х | х | Х |
| At least one serious adverse event <sup>b</sup> | X | х | х | х | х | Х |
| At least one related, serious adverse event | X | х | х | х | х | Х |
| At least one adverse event leading to early termination <sup>c</sup> | X | х | х | х | х | х |
| At least one medically attended adverse event | х | Х | х | х | х | х |

Note: N = Number of participants in the Safety Population

<sup>&</sup>lt;sup>a</sup> Participants are counted once for each category regardless of the number of events.

<sup>&</sup>lt;sup>b</sup> A listing of Serious Adverse Events is included in Section 9.3

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.

## 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

#### **Table 52:** Listing of Serious Adverse Events– Safety Population

[Implementation Note: This listing is included in the table shells document, as it is included in the body of the CSR. If the event is ongoing (no stop date), indicate "ongoing" for the "Duration". If more than one reason is selected for the reason reported as an SAE, list all reasons in the column, separated by a comma. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. If there are no comments for an event, populate 'Comments' row with 'None'. Add columns for MedDRA HLT or LLT depending on halting criteria or other study needs. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Listing should be sorted by Treatment Group, Participant ID, Associated with Dose No., and No. of Days Post Associated Dose.]

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Group: , Partic | cipant ID: , AE | Number: | | | | | | | | | |
| | l | Ι | | | | l | l | 1 | | | 1 | |
| Comments: | | | | | | L | L | | <u> </u> | | | 1 |
| Participant | t ID: , Treatme | nt Group: , AE | Number: | | | | | | | | | |
| Comments: | | | | | | | | | | | | |

**Table 53:** Listing of Non-Serious Adverse Events of Moderate or Greater Severity – Safety Population

[Implementation Note: Listing should be sorted by Treatment Group, Participant ID, Associated with Dose No., and No. of Days Post Associated Dose.]

| Adverse<br>Event | Associated<br>with Dose<br>No. | No. of<br>Days Post<br>Associated<br>Dose<br>(Duration) | No. of<br>Days Post<br>Dose the<br>Event<br>Became<br>Serious | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Group: , Parti | cipant ID: , A | E Number: | | | | | | | | |
| Comments | | | | | | | | | | | |
| Participan | t ID: , Treatme | ent Group: , A | E Number: | | | | | | | | |
| Comments | | | | | | | | | | | |

Table 54: Adverse Events Occurring in ≥ 5% of Participants in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group - Safety Population

| | MedDRA System Organ | | 4CMenB<br>(N=X) | | | Placebo<br>(N=X) | | A | All Participan<br>(N=X) | ts |
|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term | Class | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | | | | | | | | | | |
| All | All | X | X | X | X | X | X | X | х | х |
| PT1 | SOC1 | X | X | X | X | X | X | X | х | х |
| Etc. | Etc. | X | X | X | X | X | X | X | х | х |
| Other (Non-serious) Adverse Events | | | | | | | | | | |
| All | All | X | X | X | X | X | X | X | х | Х |
| PT1 | SOC1 | Х | x | X | X | X | X | x | х | х |
| Etc. | Etc. | Х | х | X | X | X | X | х | х | х |

Notes: N = number of participants in the Safety Population (number of participants at risk).

n= number of participants reporting event.

Events= total frequency of events reported.

#### 14.3.1.1 Solicited Adverse Events

Table 55: Number and Percentage of Participants Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Maximum Severity, Dose, and Treatment Group – Safety Population

| | | Post D | | 4CMenB | | • | Placebo | | | 4CMenB | Post | Dose 2 · | - Placebo | Pos | st Either<br>4CMe<br>(N=X | nB | Po | ost Eith<br>Place<br>(N= | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> |
| Any | Any Severity | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| Symptom | None | X | XX | x, x | X | xx | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| | Mild | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Moderate | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| Systemic Syr | nptoms | | | | | | | | | | | | | | | | | | |
| | Any Severity | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| Any | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| Systemic | Mild | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| Symptom | Moderate | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Any Severity | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| [Systemic<br>Symptom 1] | Mild | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Moderate | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| | Any Severity | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x |
| [Systemic<br>Symptom 2] | Mild | X | XX | x, x | X | XX | x, x | Х | XX | x, x | х | XX | x, x | Х | XX | x, x | X | xx | x, x |
| J | Moderate | X | XX | x, x | X | xx | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x | X | xx | x, x |
| | Severe | X | XX | x, x | X | xx | x, x | X | XX | x, x | X | XX | x, x | X | xx | x, x | X | xx | x, x |

Table 55: Number and Percentage of Participants Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Maximum Severity, Dose, and Treatment Group – Safety Population (continued)

| | | Post D | 0ose 1 - 4<br>(N=X) | 4CMenB | Post 1 | Dose 1 -<br>(N=X | Placebo | Post I | Oose 2 -<br>(N=X | 4CMenB | Post | Dose 2 -<br>(N=X | · Placebo | Pos | t Either<br>4CMer<br>(N=X | nB | Po | ost Eith<br>Place<br>(N= | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> | n | % | 95% CI <sup>a</sup> |
| Local Sympt | oms | | | | | | | | | | | | | | | | | | |
| | Any Severity | X | XX | x, x | X | XX | x, x | X | xx | x, x | X | xx | x, x | X | XX | x, x | X | XX | x, x |
| | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| Any Local<br>Symptom | Mild | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | x | XX | x, x |
| - 7 | Moderate | X | xx | x, x | X | XX | x, x | x | xx | x, x | X | xx | x, x | X | XX | x, x | x | xx | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| | Any Severity | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | х | XX | x, x |
| [Local<br>Symptom 1] | Mild | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| Symptom 1 | Moderate | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| [Local | Any Severity | X | XX | x, x | X | XX | x, x | x | xx | x, x | X | XX | x, x | X | XX | x, x | x | xx | x, x |
| Symptom 2] | None | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Mild | X | XX | x, x | X | XX | x, x | X | xx | x, x | Х | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Moderate | X | XX | x, x | X | XX | x, x | X | xx | x, x | Х | XX | x, x | X | XX | x, x | X | XX | x, x |
| | Severe | X | XX | x, x | X | XX | x, x | X | xx | x, x | Х | XX | x, x | X | XX | x, x | X | XX | x, x |

Note: N = Number of participants in the Safety Population who received the specified dose. Severity is the maximum severity reported over all solicited symptoms post dosing for each participant.

a The 95% CI of the proportion will be calculated using Clopper-Pearson (Exact) methodology from a binomial distribution.

Table 56: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing - 4CMenB, Post Dose 1

| | | Pre-l | Dose 1 | Post- | Dose 1 | Da | y 1 | Da | ıy 2 | Da | ıy 3 | Da | ay 4 | Da | ny 5 | Da | ny 6 | Day | y <b>7</b> + |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Symptom | None | Х | XX | х | XX | Х | XX | Х | XX | Х | XX | х | XX | х | XX | Х | XX | Х | XX |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Systemic Sympt | oms | • | • | • | | | • | | • | | • | • | • | • | • | | • | | |
| Any Systemic | None | X | XX | х | XX | X | XX | X | XX | Х | XX | X | XX | х | XX | X | XX | X | XX |
| Symptom | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic | None | | | | | | | | | | | | | | | | | | |
| Symptom 1] | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Systemic | None | | | | | | | | | | | | | | | | | | |
| Symptom 2] | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| <b>Local Symptom</b> | s | | | | | | | | | | | | | | | | | | |
| Any Local | None | Х | XX | X | XX | X | xx | X | xx | X | XX | X | XX | X | XX | X | xx | X | xx |
| Symptom | Mild | | | | | | | | | | | | | | | | | | |

Table 56: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing - 4CMenB, Post Dose 1 (continued)

| | | Pre-I | Oose 1 | Post-l | Dose 1 | Da | ıy 1 | Da | y 2 | Da | y 3 | Da | ıy 4 | Da | y 5 | Da | ıy 6 | Day | y 7+ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Local Symptom | None | | | | | | | | | | | | | | | | | | |
| 1] | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| [Local Symptom | None | | | | | | | | | | | | | | | | | | |
| 2] | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |

Note: N = Number of participants in the Safety Population who received the specified dose. Severity is the maximum severity reported post dosing for each participant for each day.

#### Tables with similar format:

- Table 57: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing- 4CMenB, Post Dose 2
- Table 58: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing- Placebo, Post Dose 1
- Table 59: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Placebo, Post Dose 2

Table 60: Number and Percentage of Participants Experiencing Solicited Events for Dose 1 Compared with Dose 2 by Treatment Group

| Treatment Group | | Dose 2 – Participants with No<br>Symptoms | Dose 2 – Participants with Mild or<br>Greater Symptoms | Dose 2 – Total Number of<br>Participants |
|---|---|---|---|---|
| Systemic Symptoms | | | | |
| | Dose 1 Participant with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Participants with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| 4CMenB | Dose 1 Total Number of Participants | x (%) | x (%) | x (100%) |
| | Dose 1 Participant with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Participants with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| Placebo | Dose 1 Total Number of Participants | x (%) | x (%) | x (100%) |
| Local Symptoms | | | | |
| | Dose 1 Participants with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Participants with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| 4CMenB | Dose 1 Total Number of Participants | x (%) | x (%) | x (100%) |
| | Dose 1 Participants with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Participants with Mild or Greater<br>Symptoms | x (%) | x (%) | x (%) |
| Placebo | Dose Total Number of Participants | x (%) | x (%) | x (100%) |

Notes: Denominators for percentages are the number of participants in the Safety Population who received both the first and second dose.

#### 14.3.1.2 Unsolicited Adverse Events

Summary of Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Dose Number, and Treatment Table 61: Group

| | | | | 4 | CMenB | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Post Do | ose 1 (N=X) | | | Post Do | se 2 (N=X) | | | Post An | y Dose (N= | X) |
| MedDRA Preferred Term | MedDRA Preferred Term | n | % | 95% CI | Events | n | % | 95% CI | Events | n | % | 95% CI | Events |
| Any SOC | Any PT | Х | XX | xx, xx | х | Х | xx | xx, xx | х | X | XX | xx, xx | x |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| | | | • | ] | Placebo | | • | • | | | 1 | | |
| MedDRA System Organ | | | Post Do | se 1 (N=X) | | | Post Do | se 2 (N=X) | | | Post An | y Dose (N= | X) |
| Class | MedDRA Preferred Term | n | % | 95% CI | Events | n | % | 95% CI | Events | n | % | 95% CI | Events |
| Any SOC | Any PT | Х | XX | xx, xx | х | Х | xx | xx, xx | х | X | XX | xx, xx | x |
| [SOC 1] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | | | |
| | [PT 1] | | | | | | | | | | | | |
| | [PT 2] | | | | | | | | | | | | |

point.

Table 62: Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Maximum Severity, Relationship, and **Treatment Group** 

| | | | | 4CMenB | | | | | | | | | ts | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA System<br>Organ Class | Preferred Term | Severity | Related | | Not<br>Related | | Total | | Related | | Not<br>Related | | Total | | Related | | Not<br>Related | | Total | |
| | | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | Any Severity | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Mild | X | XX | X | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Moderate | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Severe | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| SOC 1 | PT 1 | Any Severity | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Mild | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Moderate | X | xx | X | XX | X | XX | х | xx | х | XX | X | xx | х | xx | х | xx | х | xx |
| | | Severe | х | xx | х | XX | X | XX | х | xx | х | XX | х | xx | х | xx | х | xx | х | xx |
| | PT 2 | Any Severity | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Mild | х | XX | х | XX | X | XX | х | XX | х | XX | X | XX | х | XX | х | XX | х | XX |
| | | Moderate | х | xx | X | XX | X | XX | х | xx | х | XX | X | xx | х | xx | х | xx | х | xx |
| | | Severe | х | xx | X | XX | X | XX | х | xx | х | XX | X | xx | х | xx | х | xx | х | xx |

**Table 63:** Related Unsolicited Adverse Events Within 7 Days Post Dosing by MedDRA System Organ Class and Preferred Term, Dose, and **Treatment Group** 

[Implementation Note: Day x-y interval should correspond to period of collection for solicited symptoms, if applicable.]

| | | | | Day 1-7<br>Post Dose | 1 | | Day 1-7<br>Post Dose 2 | 2 | Within 7 | Days Post l | Either Dose |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | MedDRA System Organ Class | MedDRA Preferred Term | eferred Term n % Events n % | Events | n | % | Events | | | | |
| 4CMenB Any SOC | Any PT | X | xx | х | X | xx | х | х | xx | х | |
| $(\mathbf{N} = \mathbf{X})$ | [SOC 1] | Any PT | | | | | | | | | |
| | | [PT 1] | | | | | | | | | |
| | | [PT 2] | | | | | | | | | |
| | [SOC 2] | Any PT | | | | | | | | | |
| | | [PT 1] | | | | | | | | | |
| | | [PT 2] | | | | | | | | | |
| Placebo | Any SOC | Any PT | x | xx | x | x | XX | x | x | xx | х |
| (N=X) | [SOC 1] | Any PT | | | | | | | | | |
| | | [PT 1] | | | | | | | | | |
| | | [PT 2] | | | | | | | | | |

Note: N = Number of participants in the Safety Population. This table presents number and percentage of participants. For each time point, a participant is only counted once per PT.

 Table 64:
 Laboratory Assessment --RPR Results - Safety Population

| | Treatment | | Posi | itive | Ne | gative | Missing | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Group | N | n | % | n | % | n | % |
| Baseline | 4CMenB | х | х | XX | X | XX | Х | XX |
| | Placebo | | | | | | | |
| Day 29 | 4CMenB | | | | | | | |
| | Placebo | | | | | | | |
| Day 181 | 4CMenB | | | | | | | |
| | Placebo | | | | | | | |
| Max Severity Post | 4CMenB | | | | | | | |
| Baseline | Placebo | | | | | | | |
| Note: N = Number o | f available participa | nts in the | Safety Popula | tion at certain | time | | | |

Table 65: Laboratory Assessment --HIV Antibody Testing Results - Safety Population

| | Treatment | | Pos | itive | Neg | ative | Missing | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Group | N | n | % | n | % | n | % |
| Baseline | 4CMenB | X | X | XX | X | xx | X | XX |
| | Placebo | | | | | | | |
| Day 181 | 4CMenB | | | | | | | |
| | Placebo | | | | | | | |
| Max Severity Post | 4CMenB | | | | | | | |
| Baseline | Placebo | | | | | | | |
| Note: N = Number of | available participa | nts in the | Safety Populati | on at certain tim | ne | • | • | • |

Table 66: Laboratory Assessment – Chlamydia NAAT Testing Results - Safety Population

| Test | | | | Pos | itive | Neg | ative | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|
| | Time Point | Treatment Group | N | n | % | n | % | n | % |
| Chlamydia | Baseline | 4CMenB | х | х | xx | х | xx | х | XX |
| NAAT<br>Genitourinary | | Placebo | | | | | | | |
| ٠ | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| Chlamydia | Baseline | 4CMenB | | | | | | | |
| NAAT<br>Rectal | | Placebo | | | | | | | |
| | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| Chlamydia | Baseline | 4CMenB | | | | | | | |
| NAAT<br>Pharyngeal | | Placebo | | | | | | | |
| v 0 | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| Note: N = Num | ber of available partic | pants in the Safety Population | at certain | time | • | • | • | • | • |

**Table 67:** Laboratory Assessment – Gonorrhea NAAT Testing Results - Safety Population

| Test | | Treatment | | Pos | sitive | Neg | gative | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|
| | Time Point | Group | N | n | % | n | % | n | % |
| Gonorrhea | Baseline | 4CMenB | х | X | XX | Х | xx | х | XX |
| NAAT<br>Genitourinary | | Placebo | | | | | | | |
| | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| Gonorrhea | Baseline | 4CMenB | | | | | | | |
| NAAT<br>Rectal | | Placebo | | | | | | | |
| | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| Gonorrhea | Baseline | 4CMenB | | | | | | | |
| NAAT<br>Pharyngeal | | Placebo | | | | | | | |
| | Day 29 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |
| | Day 181 | 4CMenB | | | | | | | |
| | | Placebo | | | | | | | |

**Table 68:** Laboratory Assessment – Trichomonas Testing Results - Safety Population

| | Treatment | | Posi | itive | Neg | ative | Missing | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Group | N | n | % | n | % | n | % |
| Baseline | 4CMenB | X | Х | xx | X | xx | X | XX |
| | Placebo | | | | | | | |
| Day 29 | 4CMenB | | | | | | | |
| | Placebo | | | | | | | |
| Day 181 | 4CMenB | | | | | | | |
| | Placebo | | | | | | | |
| Note: N = Number o | f available participar | ts in th | e Safety Populat | ion at certain tin | ne. | | | • |

Table 69: Number and Percentage of Participants with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group

| WHO Drug Code<br>Level 1, Anatomic Group | WHO Drug Code<br>Level 2, Therapeutic | | MenB<br>N=X) | | cebo<br>(=X) | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|
| | Subgroup | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | XX | Х | xx | x | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | |
| | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |
| | [ATC 2 - 3] | | | | | | |
| [ATC Level 1 – 2] | Any [ATC 1 – 2] | | | | | | |
| | [ATC 2 - 1] | | | | | | |
| | [ATC 2 - 2] | | | | | | |

Note: N = Number of participants in each group in the Safety Population.

n = Number of participants reporting taking at least one medication in the specific WHO Drug Class.

# **APPENDIX 2. FIGURE MOCK-UPS**

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram- Disposition of Participants |
|---|---|
| Figure 2: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 3: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day,<br>Sex and Treatment Group - Immunogenicity Population |
| Figure 4: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 5: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day,<br>Sex and Treatment Group - Per-Protocol Population |
| Figure 6: | Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 7: | Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day, Sex and Treatment Group - Immunogenicity Population |
| Figure 8: | Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 9: | Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day, Sex and Treatment Group - Per-Protocol Population |
| Figure 10: | Geometric Mean Titers of Serum IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 11: | Geometric Mean Titers of Serum IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 12: | Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 13: | Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 14: | Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against OMV by Study<br>Day and Treatment Group - Immunogenicity Population |
| Figure 15: | Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against OMV by Study<br>Day and Treatment Group - Per-Protocol Population |
| Figure 16: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 17: | Geometric Mean Titers of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |

| Figure 18: | Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
|---|---|
| Figure 19: | Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 20: | Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 21: | Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 22: | Geometric Mean Titers of Serum IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 23: | Geometric Mean Titers of Serum IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 24: | Geometric Mean Titers of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 25: | Geometric Mean Titers of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 26: | Geometric Mean Titers of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 27: | Geometric Mean Titers of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 28: | Geometric Mean Titers of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 29: | Geometric Mean Titers of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 30: | Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 31: | Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 32: | Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 33: | Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 34: | Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 35: | Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 36: | Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population116 |
|---|---|
| Figure 37: | Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 38: | Titers of Serum Bactericidal Antibody Against by Study Day and Treatment Group - Immunogenicity Population |
| Figure 39: | Titers of Serum Bactericidal Antibody Against by Study Day and Treatment Group - Per-Protocol Population |
| Figure 40: | Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 41: | Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against OMV by Day and Treatment Group - Per-Protocol Population |
| Figure 42: | Reverse Cumulative Distribution of Serum IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 43: | Reverse Cumulative Distribution of Serum IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 44: | Reverse Cumulative Distribution of Serum IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 45: | Reverse Cumulative Distribution of Serum IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 46: | Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 47: | Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 48: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 49: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 50: | Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 51: | Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 52: | Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 53: | Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |

| Figure 54: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population118 |
|---|---|
| Figure 55: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population118 |
| Figure 56: | Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 57: | Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 58: | Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 59: | Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 60: | Reverse Cumulative Distribution of Serum IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 61: | Reverse Cumulative Distribution of Serum IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 62: | Reverse Cumulative Distribution of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 63: | Reverse Cumulative Distribution of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 64: | Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population |
| Figure 65: | Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population |
| Figure 66: | Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population |
| Figure 67: | Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population |
| Figure 68: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population119 |
| Figure 69: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population119 |
| Figure 70: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population119 |
| Figure 71: | Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against NHBAby Study Day and Treatment Group - Per-Protocol Population119 |

| Figure 72: | Reverse Cumulative Distribution of Serum Bactericidal Antibody Against GC Study Day and Treatment Group - Immunogenicity Population |
|---|---|
| Figure 73: | Reverse Cumulative Distribution of Serum Bactericidal Antibody Against GC by Study Day and Treatment Group - Per-Protocol Population |
| Figure 74: | Frequencies and Function of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population120 |
| Figure 75: | Frequencies and Function of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population |
| Figure 76: | Frequencies and Function of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group - Immunogenicity Population |
| Figure 77: | Frequencies and Function of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group - Per-Protocol Population |
| Figure 78: | Frequencies and Function of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population |
| Figure 79: | Frequencies and Function of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population |
| Figure 80: | Frequencies and Function of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population120 |
| Figure 81: | Frequencies and Function of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population120 |
| Figure 82: | Frequencies and Function of Peripheral Blood CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population120 |
| Figure 83: | Frequencies and Function of Peripheral Blood CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population120 |
| Figure 84: | Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population120 |
| Figure 85: | Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population121 |
| Figure 86: | Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population121 |
| Figure 87: | Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Per-Protocol Population121 |
| Figure 88: | Number and Severity of Adverse Events by MedDRA System Organ Class and Treatment Group |
| Figure 89: | Maximum Severity of Solicited Events by Reaction and Treatment Group123 |
| Figure 90: | Maximum Severity of Solicited Events per Participant by Days Post Treatment and Treatment Group |

| Figure 91: | Number of Adverse Events by MedDRA System Organ Class and Severity125 |
|---|---|
| Figure 92: | Number of and Percentage of Participants Experiencing Adverse Events by MedDRA System Organ Class and Maximum Severity |
| Figure 93: | Number of Adverse Events by MedDRA System Organ Class and Relationship to Treatment |
| Figure 94: | Number of and Percentage of Participants Experiencing Adverse Events by MedDRA System Organ Class and Relationship to Treatment |

Figure 1: CONSORT Flow Diagram- Disposition of Participants



# Figure 2: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population

[Implementation Note: A generic sample figure is shown below. Planned study day is plotted along the x-axis, with visit labels as tick labels. Titer/frequency is plotted on the y-axis. Separated panels will be used for different antigens- Ng1291 and CNG20. Different colors indicate different treatment groups and/or sex. Scale will be determined for each antigen separately based on the distribution of the data received). GMT/frequency will be plotted at each visit with upper and lower error bars for the 95% CI for each study arm with different marker shapes/colors for each study arm.]



Figures with similar format (for Serum, include NZ98, Ng1291 and CNG20; For mucosal, only include Ng1291 and CNG20.):

- Figure 3: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day, Sex and Treatment Group Immunogenicity Population
- Figure 4: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 5: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against OMV by Study Day, Sex and Treatment Group - Per-Protocol Population
- Figure 6: Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 7: Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day, Sex and Treatment Group Immunogenicity Population
- Figure 8: Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 9: Geometric Mean Titers of Serum IgG Antibody Against OMV by Study Day, Sex and Treatment Group Per-Protocol Population

- Figure 10: Geometric Mean Titers of Serum IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 11: Geometric Mean Titers of Serum IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 12: Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 13: Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 14: Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 15: Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population

Following analysis (Figure 16-21) will be performed based on the results of the interim analysis and specimen availability

- Figure 16: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 17: Geometric Mean Titers of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 18: Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 19: Geometric Mean Titers of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 20: Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 21: Geometric Mean Titers of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 22: Geometric Mean Titers of Serum IgA Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 23: Geometric Mean Titers of Serum IgA Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 24: Geometric Mean Titers of Serum IgA Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 25: Geometric Mean Titers of Serum IgA Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 26: Geometric Mean Titers of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population

**Per-Protocol Population** 

Geometric Mean Titers of Rectal Mucosal IgA Antibody Against OMV by Study Day and Figure 27: **Treatment Group - Per-Protocol Population** Geometric Mean Titers of Rectal Mucosal IgA Antibody Against NHBA by Study Day Figure 28: and Treatment Group - Immunogenicity Population Figure 29: Geometric Mean Titers of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population Figure 30: Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population Figure 31: Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population Figure 32: Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population Geometric Mean Titers of Vaginal Mucosal IgA Antibody Against NHBA by Study Day Figure 33: and Treatment Group - Per-Protocol Population Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Figure 34: Day and Treatment Group - Immunogenicity Population Figure 35: Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population Figure 36: Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population Geometric Mean Titers of Oropharyngeal Mucosal IgA Antibody Against NHBA by Figure 37: Study Day and Treatment Group - Per-Protocol Population Figure 38: Titers of Serum Bactericidal Antibody Against by Study Day and Treatment Group -**Immunogenicity Population** Figure 39: Titers of Serum Bactericidal Antibody Against by Study Day and Treatment Group -

Figure 40: Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population

[Implementation Note: An example figure is shown below. The figures for each antigen (OMV98, OMV1291, and OMV20) will have one column with time points (Day 1, Day 15, Day 29, Day 43, Day 57, Day 181). There will be 3x6 panels in this figure. Study arms will be plotted with different marker/line colors.]



Figures with similar format:

Figure 41: Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against OMV by Day and Treatment Group - Per-Protocol Population

Figure 42: Reverse Cumulative Distribution of Serum IgG Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population

- Figure 43: Reverse Cumulative Distribution of Serum IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 44: Reverse Cumulative Distribution of Serum IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 45: Reverse Cumulative Distribution of Serum IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 46: Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 47: Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 48: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 49: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population

Following analysis (Figure 50-73) will be performed based on the results of the interim analysis and specimen availability

- Figure 50: Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 51: Reverse Cumulative Distribution of Rectal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 52: Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 53: Reverse Cumulative Distribution of Vaginal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 54: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population
- Figure 55: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgG Antibody Against NHBA by Study Day and Treatment Group Per-Protocol Population
- Figure 56: Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group Immunogenicity Population
- Figure 57: Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group Per-Protocol Population
- Figure 58: Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group Immunogenicity Population

Figure 73:

Reverse Cumulative Distribution of Rectal Mucosal IgA Antibody Against NHBA by Figure 59: Study Day and Treatment Group - Per-Protocol Population Reverse Cumulative Distribution of Serum IgA Antibody Against OMV by Study Day Figure 60: and Treatment Group - Immunogenicity Population Figure 61: Reverse Cumulative Distribution of Serum IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population Figure 62: Reverse Cumulative Distribution of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population Figure 63: Reverse Cumulative Distribution of Serum IgA Antibody Against NHBA by Study Day and Treatment Group - Per-Protocol Population Figure 64: Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population Figure 65: Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against NHBA by Figure 66: Study Day and Treatment Group - Immunogenicity Population Reverse Cumulative Distribution of Vaginal Mucosal IgA Antibody Against NHBA by Figure 67: Study Day and Treatment Group - Per-Protocol Population Figure 68: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Immunogenicity Population Figure 69: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against OMV by Study Day and Treatment Group - Per-Protocol Population Figure 70: Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against NHBA by Study Day and Treatment Group - Immunogenicity Population Reverse Cumulative Distribution of Oropharyngeal Mucosal IgA Antibody Against Figure 71: NHBAby Study Day and Treatment Group - Per-Protocol Population Figure 72: Reverse Cumulative Distribution of Serum Bactericidal Antibody Against GC Study Day and Treatment Group - Immunogenicity Population

Reverse Cumulative Distribution of Serum Bactericidal Antibody Against GC by Study

Day and Treatment Group - Per-Protocol Population

Figure 74: Frequencies and Function of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group - Immunogenicity Population

[Implementation Note: A generic sample figure is shown below. Planned study day is plotted along the x-axis, with visit labels as tick labels. Titer/frequency is plotted on the y-axis (Scale will be determined for NZ98, Ng1291 and CNG20 from OMV or NHBA separately based on the distribution of the data received). Frequency will be plotted at each visit with upper and lower error bars for the 95% CI for each study arm with different marker shapes/colors for each study arm.]



Figures with similar format:

- Figure 75: Frequencies and Function of Memory B Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 76: Frequencies and Function of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group Immunogenicity Population
- Figure 77: Frequencies and Function of Peripheral Blood T Cells Specific for OMV Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 78: Frequencies and Function of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group Immunogenicity Population
- Figure 79: Frequencies and Function of Peripheral Blood T Cells Specific for NHBA Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 80: Frequencies and Function of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Immunogenicity Population
- Figure 81: Frequencies and Function of Peripheral Blood CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 82: Frequencies and Function of Peripheral Blood CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Immunogenicity Population
- Figure 83: Frequencies and Function of Peripheral Blood CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 84: Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Immunogenicity Population

- Figure 85: Frequencies and Function of Rectal Mucosal CD4+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Per-Protocol Population
- Figure 86: Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Immunogenicity Population
- Figure 87: Frequencies and Function of Rectal Mucosal CD8+ T Cells Specific for OMV and NHBA Antigens by Time Point and Treatment Group Per-Protocol Population

Figure 88: Number and Severity of Adverse Events by MedDRA System Organ Class and Treatment Group





Figure 89: Maximum Severity of Solicited Events by Reaction and Treatment Group

Figure 90: Maximum Severity of Solicited Events per Participant by Days Post Treatment and Treatment Group







Figure 92: Number of and Percentage of Participants Experiencing Adverse Events by MedDRA System Organ Class and Maximum Severity

[Implementation Note: This figure includes serious and non-serious unsolicited adverse events deemed related to study product. The SOCs should be sorted in descending incidence; e.g., for this figure, "Infections and infestations" should be listed first.]



Figure 93: Number of Adverse Events by MedDRA System Organ Class and Relationship to Treatment



Figure 94: Number of and Percentage of Participants Experiencing Adverse Events by MedDRA System Organ Class and Relationship to Treatment



## APPENDIX 3. LISTINGS MOCK-UPS

### LISTINGS

| Listing 1: | Participants Receiving Investigational Product |
|---|---|
| Listing 2: | Early Terminations or Discontinued Participants |
| Listing 3: | Participant-Specific Protocol Deviations |
| Listing 4: | Non-Participant-Specific Protocol Deviations |
| Listing 5: | Participants Excluded from Analysis Populations |
| Listing 6: | Demographic Data |
| Listing 7: | Pre-Existing and Concurrent Medical Conditions |
| Listing 8: | Treatment Compliance Data |
| Listing 9: | Immunogenicity Response Data ELISA– Rectal Mucosal |
| Listing 10: | Immunogenicity Response Data ELISA – Serum against OMV and NHBA antigens139 |
| Listing 11: | Immunogenicity Response Data ELISA – Vaginal Mucosal against OMV and NHBA antigens |
| Listing 12: | Immunogenicity Response Data ELISA – Oropharyngeal Mucosal against OMV and NHBA antigens |
| Listing 13: | Immunogenicity Response Data ELISA – Serum Bactericidal against N. gonorrhoeae139 |
| Listing 14: | Immunogenicity Response Data ELISA – Serum Bactericidal against N. meningitidis139 |
| Listing 15: | Immunogenicity Response Data -Frequencies of Immuno-cells Specific for OMV Antigens- ELISpot |
| Listing 16: | Immunogenicity Response Data -Frequencies of Immuno-cells Specific for NHBA Antigens - ELISpot |
| Listing 17: | Immunogenicity Response Data - Frequencies of Peripheral Blood T cells Specific142 |
| Listing 18: | Immunogenicity Response Data – Frequencies of Peripheral Blood CD4+ T Cells Specific for Antigens - ICS |
| Listing 19: | Immunogenicity Response Data – Frequencies of Peripheral Blood CD8+ T Cells Specific for Antigens– ICS |
| Listing 20: | Immunogenicity Response Data – Frequencies of Rectal Mucosal CD4+ T Cells Specific for Antigens– ICS |
| Listing 21: | Immunogenicity Response Data – Frequencies of Rectal Mucosal CD8+ T Cells Specific for Antigens– ICS |
| Listing 22: | Immunogenicity Response Data – Gonococcal Adhesion to Human Cervical Cell Line (ME180) by Mucosal Antibodies at Day 43 |
| Listing 23: | Solicited Events – Systemic Symptoms |

## Table of Listings (continued)

| Listing 24: Solicited Events – Local Symptoms | 146 |
|---|---|
| Listing 25: Listing of Unsolicited Adverse Events | 147 |
| Listing 26: Listing of Laboratory Assessment – Serology – Safety Population | 148 |
| Listing 27: Listing of Laboratory Assessment – STI Testing – Safety Population | 149 |
| Listing 28: Abnormal Laboratory Result - Hematology – Safety Population | 150 |
| Listing 29: Abnormal Laboratory Result - Coagulation - Enrolled Participants | 150 |
| Listing 30: Abnormal Vital Sign Findings | 151 |
| Listing 31: Abnormal Physical Exam Findings | 152 |
| Listing 32: Concomitant Medications | 153 |
| Listing 33: Pregnancy Reports – Maternal Information | 154 |
| Listing 34: Pregnancy Reports – Gravida and Para | 155 |
| Listing 35: Pregnancy Reports – Live Birth Outcomes | 156 |
| Listing 36: Pregnancy Reports – Still Birth Outcomes | 157 |
| Listing 37: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 158 |

#### **Listing 1: Participants Receiving Investigational Product**

| Treatment Group | Participant ID | Product Received Study Vaccination 1 | Product Received Study Vaccination 2 |
|---|---|---|---|

#### **Listing 2:** Early Terminations or Discontinued Participants

[Implementation Note: Category will be either "Early Termination" or "Treatment Discontinuation." In the "Reason" column, concatenate any "specify" fields, including AE number and DV number. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, alphabetically by Category (in the case a participant both terminates early and discontinues treatment).]

| Treatment Group | Participant ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|
| Note Participants who | early terminated or discontinu | ed due to Covid 10 are | nighlighted with yellow color code | |

Note. Participants who early terminated or discontinued due to Covid-19 are highlighted with yellow color code.

#### **Listing 3: Participant-Specific Protocol Deviations**

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Participant refusal." In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, DV Number.]

| Treatment<br>Group | Participant<br>ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Participant<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note. Participants who had a protocol deviation due to Covid-19 are highlighted with yellow color code.

#### **Listing 4:** Non-Participant-Specific Protocol Deviations

[Implementation Note: In the "Deviation" column, concatenate any and all "specify" fields (including visit number, etc.). If "Reason for Deviation" is "Other," concatenate "specify" field, separate by a colon, e.g., "Other: Participant refusal." Sort order: Site, Start Date.]

| Site | Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Participant<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|
| | | t- C: 1 10 1:- | | | | | | | |

Note. Protocol deviations due to Covid-19 are highlighted with yellow color code.

#### **Listing 5:** Participants Excluded from Analysis Populations

[Implementation Note: This data in this listing should be congruent with the "Analysis Populations by Treatment Group" table. The reasons included here should match the SAP text that describes who will be excluded from analyses. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification.] Sort order: Treatment Group, Participant ID.]

| Treatment Group | Participant ID | Analyses in which<br>Participant is Included | Analyses from which Participant is Excluded | Results Available? | Reason Participant Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, immunogenicity, PP] | [e.g., Safety, , immunogenicity, PP] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

#### **Listing 6:** Demographic Data

[Implementation Note: If a participant is multi-racial, in "Race" column, note "Multiple: (list races, separated by a comma)."

In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification.] Sort order: Treatment Group, Participant ID.]

| Treatment Group | Participant ID | Sex | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|

#### **Listing 7: Pre-Existing and Concurrent Medical Conditions**

[Implementation Note: "Condition Start Day" and "Condition End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). Rather than use exact study days, categorize as follows:

- 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment
- Within 1 month of enrollment
- During study
- If ongoing, display "Ongoing" in the "Condition End Day" column
- Within 1 month of enrollment
- During study
- If ongoing, display "Ongoing" in the "Condition End Day" column

It may be appropriate to add another category, based on exclusion criteria that restrict conditions within a particular time period (e.g., within 3 years prior to enrollment). In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, MH Number.]

| Treatment<br>Group | Participant<br>ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

## **Listing 8:** Treatment Compliance Data

| Treatment<br>Group | Participant<br>ID | Dose Number | Planned Study Days | Actual Study Days Administered | Compliant or Non-compliant |
|---|---|---|---|---|---|
| | | | | | Yes/No-Compliant / Non-compliant |

#### Listing 9: Immunogenicity Response Data ELISA– Rectal Mucosal

[Implementation Note: Update as appropriate for your study assay/strain and endpoints. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification.] Listing should be sorted by Treatment Group, Participant ID, Planned Time Point.]

| Treatment | | Planned | Actual Study | IgG T | iter | IgA Titer | |
|---|---|---|---|---|---|---|---|
| Group | Participant ID | Time Point | Day | OMV Ng1291 | OMV CNG20 | OMV Ng1291 | OMV CNG20 |

Listings with similar format: (for Serum specimens, include NZ98, Ng1291 and CNG20, for mucosal specimens, only include Ng1291 and CNG20)

- Listing 10: Immunogenicity Response Data ELISA Serum against OMV and NHBA antigens
- Listing 11: Immunogenicity Response Data ELISA Vaginal Mucosal against OMV and NHBA antigens
- Listing 12: Immunogenicity Response Data ELISA Oropharyngeal Mucosal against OMV and NHBA antigens
- Listing 13: Immunogenicity Response Data ELISA Serum Bactericidal against N. gonorrhoeae
- Listing 14: Immunogenicity Response Data ELISA Serum Bactericidal against N. meningitidis

Listing 15: Immunogenicity Response Data -Frequencies of Immuno-cells Specific for OMV Antigens- ELISpot

| Treatment 1 | Particinant | Planned | Actual Study | | Memory B cells | | Peripheral blood T cells | | |
|---|---|---|---|---|---|---|---|---|---|
| Group | | Time Point | Day | NZ98 OMV | Ng1291 OMV | CNG20 OMV | IFNg NZ98 OMV | IFNg 1291 OMV | IFNg CNG20 OMV |

Listing 16: Immunogenicity Response Data -Frequencies of Immuno-cells Specific for NHBA Antigens - ELISpot

| | | | | | Memory B cells | | Peripheral blood T cells | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Participant<br>ID | Planned<br>Time Point | Actual Study<br>Day | NZ98 NHBA | 1291 NHBA | CNG20 NHBA | NZ98 NHBA<br>peptide pool | 1291 NHBA peptide<br>pool | CNG20 NHBA peptide pool |

Listing 17: Immunogenicity Response Data - Frequencies of Peripheral Blood T cells Specific

| Treatment | - | Planned | Actual Study | Memory B cells | | | Peripheral blood T cells | | |
|---|---|---|---|---|---|---|---|---|---|
| Group | | Time Point | Day | NZ98 OMV | 1291 OMV | CNG20 OMV | NZ98 NHBA | 1291 NHBA | CNG20 NHBA |

Listing 18: Immunogenicity Response Data – Frequencies of Peripheral Blood CD4+ T Cells Specific for Antigens - ICS

| | Planned<br>nt Time<br>Point | Planned | Planned | Planned | Actual | | NZ98 OMV | | | Ng1291 OMV | | CNG20 OMV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | | Study<br>Day | IL17+ as a % of<br>CD4+ | TNFa+ as a % of CD4+ | IFNG+ as a % of CD4+ | IL17+ as a %<br>of CD4+ | TNFa+ as a % of CD4+ | IFNG+ as a % of CD4+ | IL17+ as a % of CD4+ | TNFa+ as a % of CD4+ | IFNG+ as a % of CD4+ | |
| | | | | _ | | | | | _ | | | |

Listings with similar format:

Listing 19: Immunogenicity Response Data – Frequencies of Peripheral Blood CD8+ T Cells Specific for Antigens– ICS

Listing 20: Immunogenicity Response Data – Frequencies of Rectal Mucosal CD4+ T Cells Specific for Antigens– ICS

Listing 21: Immunogenicity Response Data – Frequencies of Rectal Mucosal CD8+ T Cells Specific for Antigens– ICS

Listing 22: Immunogenicity Response Data – Gonococcal Adhesion to Human Cervical Cell Line (ME180) by Mucosal Antibodies at Day 43

| | | | | Percent inhibition (%) | | |
|---|---|---|---|---|---|---|
| Treatment Group | Participant ID | Planned Time Point | Actual Study Day | BAA_98 | BAA_1291 | BAA_20 |
## **Listing 23:** Solicited Events – Systemic Symptoms

[Implementation Note: This listing is not color-coded. To indicate severity for quantitative symptoms (e.g., temperature, measurements), include the grade in parentheses after the number, e.g., 100.7 (Mild). This listing includes baseline assessments in addition to post-treatment assessments. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, Dose Number, Post Dose Day, Symptom.]

| Treatment<br>Group | Participant ID | Dose Number | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

Note:

<sup>&</sup>lt;sup>a</sup> Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

MA = Data reported by participant on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

## **Listing 24:** Solicited Events – Local Symptoms

[Implementation Note: This listing is not color-coded. To indicate severity for quantitative symptoms (e.g., temperature, measurements), include the grade in parentheses after the number, e.g., 100.7 (Mild). We are not indicating the "side" or arm assessed. If the arm assessed was wrong (not the arm that received treatment), then note this error in a footnote to the listing. This listing includes baseline assessments in addition to post-treatment assessments. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, Dose Number, Post Dose Day, Symptom.]

| Treatment Group | Participant ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by participant on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

## **Listing 25:** Listing of Unsolicited Adverse Events

[Implementation Note: If the event is ongoing (no stop date), indicate "ongoing" in the "Duration" column. In the "If Not Related, Alternate Etiology" column, merge the 2 data fields for collecting alternate etiology, separate by a colon. This listing includes all unsolicited adverse events. If there are no comments for an event, populate 'Comments' row with 'None'. Add columns for MedDRA HLT or LLT depending on halting criteria or other study needs. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, Associated with Dose No., No. of Days Post Associated Dose. If the table will be multi-page, move the footnote/explanation to the footer so that it repeats for each page of the table.]

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term | MAAE<br>(Yes/No) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatmen | t Group: , Parti | cipant ID: , A | E Number: | | | | | | | | | |
| Comments | s: | | | | | | | | | | | |
| Treatmen | t Group: , Parti | icipant ID: , A | E Number: | | | | | | | | | |
| Comments | s: | | | • | | • | | • | • | | | |
| Note: For | additional deta | ails about SA | Es, see Table 52 | 2. | | | | | | | | |

# **Listing 26:** Listing of Laboratory Assessment – Serology – Safety Population

| Treatment Group | Participant ID | Planned Time Point | Actual Study Day | RPR Results | HIV Antibody |
|---|---|---|---|---|---|
| | | | | Negative/Positive/Missing | Negative/Positive/Missing |
| | | | | Negative/Positive/Missing | Negative/Positive/Missing |
| | | | | Negative/Positive/Missing | Negative/Positive/Missing |

**Listing 27:** Listing of Laboratory Assessment – STI Testing – Safety Population

| Treatment<br>Group | Participant<br>ID | Planned<br>Time Point | Actual<br>Study Day | Chlamydia<br>NAAT<br>Genitourinary | Chlamydia<br>NAAT<br>Rectal | Chlamydia<br>NAAT<br>Pharyngeal | Gonorrhea<br>NAAT<br>Genitourinary | Gonorrhea<br>NAAT<br>Rectal | Gonorrhea<br>NAAT<br>Pharyngeal | Trichomonas |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing |
| | | | | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing | Negative/<br>Positive/ Missing |

**Listing 28:** Abnormal Laboratory Result - Hematology - Safety Population

| Participant<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Participant Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Listing with similar format:

**Listing 29:** Abnormal Laboratory Result - Coagulation - Enrolled Participants

## **Listing 30:** Abnormal Vital Sign Findings

[Implementation Note: This listing includes all vital sign assessments, scheduled and unscheduled. These listings are not color-coded, but the severity should be included in parentheses after the result for abnormal assessments, e.g., 100.7 (Mild). In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, Planned Time Point.]

| Treatment<br>Group | Participant ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°F) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) | Respiratory Rate<br>(breaths/min) | Weight (kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|---|

## **Listing 31: Abnormal Physical Exam Findings**

[Implementation Note: This listing includes all physical exam findings, scheduled and unscheduled. If a participant does not have any findings upon examination, they will not be included in this listing. If reported as an AE, display "Yes" with the AE Number in parentheses, e.g., "Yes (7)". In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification.] Sort order: Treatment Group, Participant ID, Planned Time Point.]

| Treatment<br>Group | Participant ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

## **Listing 32:** Concomitant Medications

[Implementation Note: "Medication Start Day" and "Medication End Day" are relative to enrollment (which is Day 1, day before enrollment is Day -1). For medication start dates that are > 30 days prior to enrollment, rather than use exact study days, categorize as follows:

- 5 years prior to enrollment
- 1-5 years prior to enrollment
- 1-12 months prior to enrollment

If ongoing, display "Ongoing" in the "Medication End Day" column. If taken for an AE or MH, display "Yes" with the AE or MH Number in parentheses, e.g., "Yes (7)". In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, and CM Number.]

| Treatment<br>Group | Participant<br>ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

## **Listing 33:** Pregnancy Reports – Maternal Information

[Implementation Note: Only include the "Pregnancy Number" column if a participant has more than 1 pregnancy. Date of Conception will be calculated based on estimated delivery date. BMI will be calculated based on pre-pregnancy height and weight. Mother's weight gain will be calculated based on pre-pregnancy weight and end of pregnancy weight. If a major congenital anomaly with previous pregnancy, display "Yes" and the text from the "specify" field, separated by a colon. If any substance use is reported, include a listing of substance use. If autopsy revealed an alternate etiology, display "Yes" and the text from the "specify" field, separated by a colon. If abnormality in product of conception, display "Yes" and the text from the "specify" field, separated by a colon. In the CSR, Participant ID should be USUBJID (not PATID) for purposes of de-identification. Sort order: Treatment Group, Participant ID, Pregnancy Number.]

| Treatment<br>Group | Participant<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 34: Pregnancy Reports - Gravida and Para

| | | | | | | Live Births | S | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Participant<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not. <sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

**Listing 35:** Pregnancy Reports – Live Birth Outcomes

| Participant<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

# **Listing 36:** Pregnancy Reports – Still Birth Outcomes

| Participant<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

# **Listing 37:** Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Participant<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|